CLINICAL TRIAL: NCT01725126
Title: A Double-blind [Sponsor Unblinded], Randomized, Placebo-controlled, Staggered-parallel Study to Investigate the Safety, Tolerability, and Pharmacodynamics of GSK2890457 in Healthy Volunteers and Subjects With Type 2 Diabetes
Brief Title: To Investigate the Safety, Tolerability and Pharmacodynamics of GSK2890457 in Healthy Volunteers and Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116623
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: metformin; diabetes; obesity; liraglutide
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Metformin; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A - GSK2890457 (Experimental): Subjects will titrate up from a maximially tolerated dose over a 7-day period. Treatment Period is 6 weeks
  Interventions: Drug: GSK2890457; Drug: Metformin
- Part B - GSK2890457 + Liraglutide (Experimental): Subjects will titrate up from a maximially tolerated dose over a 7-day period. Treatment Period is 6 weeks
  Interventions: Drug: GSK2890457; Drug: Liraglutide
- Part C - GSK2890457 + Metformin (Experimental): Subjects will titrate up from a maximially tolerated dose over a 7-day period. Treatment Period is 6 weeks
  Interventions: Drug: GSK2890457; Drug: Metformin
- Part A - Placebo (Placebo Comparator): Subjects will titrate up from a maximially tolerated dose over a 7-day period. Treatment Period is 6 weeks
  Interventions: Drug: Placebo
- Part B - Placebo (Placebo Comparator): Subjects will titrate up from a maximially tolerated dose over a 7-day period. Treatment Period is 6 weeks
  Interventions: Drug: Placebo
- Part C - Placebo (Placebo Comparator): Subjects will titrate up from a maximially tolerated dose over a 7-day period. Treatment Period is 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2890457 — Provided as powder and capsule.
  Arms: Part A - GSK2890457; Part B - GSK2890457 + Liraglutide; Part C - GSK2890457 + Metformin
Drug: Metformin — Tablet
  Part A: Single doses on Day 1 and Day 42 orally
  Part B: Subject continues usual metformin dose through Run-in, and resumes after Treatment Period completed
  Part C: Subject continues usual metformin dose throughout study
  Arms: Part A - GSK2890457; Part C - GSK2890457 + Metformin
Drug: Placebo — Provided as powder and Capsule.
  Arms: Part A - Placebo; Part B - Placebo; Part C - Placebo
Drug: Liraglutide — Provided as Injection. 6mg/mL, 3mL injector pen that permits doses of 0.6mg, 1.2mg, and 1.8mg
  Subcutaneous injection 18 weeks dosing (Stabilization and Treatment Periods, Part B only
  Other Names: Victoza
  Arms: Part B - GSK2890457 + Liraglutide

SUMMARY:
This study is the first administration of GSK2890457 in humans. The study will be conducted in 3 parts: - Part A (conducted at a single investigative site) will determine the safety and tolerability of GSK2890457 alone in healthy subjects during six weeks of dosing, as well as evaluating the potential for a pharmacokinetic interaction with metformin. Part A consists of Screening, Treatment (6 weeks) and Follow-up periods. - Part B (conducted at multiple sites) will determine safety, tolerability, and pharmacodynamics (PD) in subjects with Type 2 diabetes (T2D) when co-dosed for six weeks with liraglutide (Victoza). Part B consists of Screening, Run-in (1 week), Stabilization (12 weeks), Treatment (6 weeks) and Follow-up periods. - Part C (conducted at multiple sites) will determine safety, tolerability, and PD in subjects with T2D when co-dosed for 6 weeks with metformin. Part C consists of Screening, Run-in (1 week), Stabilization (12 weeks), Treatment (6 weeks) and Follow-up periods.

ELIGIBILITY:
Inclusion Criteria:Part A (Healthy Subjects)

* Subject able to understand and voluntarily provide the consent to participate in the study
* 18 - 70 years of age, inclusive, at the time of signing the informed consent and Body Mass Index (BMI) between 18.0 and 35.0 Kilogram (kg) per m^2, inclusive
* Understands and is willing, able and likely to be compliant with taking study drug and comply with all study procedures and restrictions
* Subject is willing to consume the foods that are part of the standardized breakfast, lunch, and dinner
* In good general health with no clinically significant and relevant abnormalities of medical history or physical examination which includes adequate renal function, alanine transaminase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper Limit of Normal (ULN )
* QTcF < 450 millisecond (msec); or QTcF < 480msec for subjects with right Bundle Branch Block
* Females must be post-menopausal
* Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment
* Females who are > 3 months postpartum and who have undergone a surgical sterilization procedure are eligible to participate in consultation with the GSK Medical Monitor

Parts B and C (Type 2 Diabetic Subjects)

* All the criteria mentioned in Part A except Body Mass Index (BMI) should be between 30.0 and 42.0 kg per m^2
* Diagnosis of T2D for at least 3 months, as defined by the American Diabetes Association
* All T2D subjects must meet label recommendations for metformin
* For Part B, subjects must be willing to discontinue metformin and replace it with daily liraglutide administered by subcutaneous injection and they must meet label recommendations
* No personal history or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia syndrome type 2

Exclusion Criteria:

* History of gastrointestinal disease, current or chronic history of liver disease, history of serious, severe or unstable physical or psychiatric illness , significant cardiovascular disease, surgery for weight loss or gastrointestinal surgery within 3 months of screening, any documented or reported eating disorder, uncontrolled hypertension, as evidenced by systolic pressure>160 or diastolic pressure >90 mmHg
* Positive test for HIV, Hepatitis B, or Hepatitis C at Screening
* Subjects with significant ECG abnormalities
* For subjects in Part C (continuing metformin), history of untreated pernicious anemia or who have laboratory parameters suggestive of subclinical megaloblastic anemia
* Presence of or symptoms of an active infection
* Uncorrected Thyroid Dysfunction
* History of chronic or acute pancreatitis
* Currently dieting to lose weight including, but not limited to, participation in a program designed to alter body weight within the last 60 days and unwilling to maintain relatively consistent exercise patterns throughout the study
* Current or recent history (within one year of screening) of alcohol or other substance abuse
* Unable to refrain from the use of non-prescription drugs
* Current participation in another clinical study or participation in a clinical study involving an investigational drug within 30 days of the screening visit
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-02-10 (Actual); Primary Completion 2013-09-12 (Actual); Study Completion 2013-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hodge RJ, Paulik MA, Walker A, Boucheron JA, McMullen SL, Gillmor DS, Nunez DJ. Weight and Glucose Reduction Observed with a Combination of Nutritional Agents in Rodent Models Does Not Translate to Humans in a Randomized Clinical Trial with Healthy Volunteers and Subjects with Type 2 Diabetes. PLoS One. 2016 Apr 19;11(4):e0153151. doi: 10.1371/journal.pone.0153151. eCollection 2016. PMID 27093610
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116623 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 3 parts in healthy male and female participants aged 18 to 70 years in Part A and in participants with type 2 diabetes (T2D) in Part B and C across three centers of United States of America.
Pre-assignment Details: A total of 15 participants were randomized in Part A, 20 were randomized in Part B and 18 were randomized in Part C.
Groups:
- Part A-Placebo: Healthy participants received oral dose of matching placebo to GSK2890457 as units of 5 gram (g) kit twice daily (BID) for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 milliliter (mL) of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) prior to breakfast (morning) and 10 g (2 unit) prior to dinner (evening). On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. On Day 1 and 42, after overnight fasting, participants received 500 milligram (mg) immediate release (IR) tablet of metformin just before breakfast. On Day 1 (5 g) and Day 42, matching placebo to GSK2890457 was given in the evening.
- Part A-GSK2890457: Healthy participants received oral dose of GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. On Day 1 and 42, after overnight fasting, participants received 500 mg IR tablet of metformin just before breakfast. On Day 1 (5 g) and Day 42, GSK2890457 was given in the evening.
- Part B-Placebo+Liraglutide: Participants with T2D, received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. Participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2, dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants received liraglutide up to 1.8 milligram (mg) once daily by subcutaneous injection during the Treatment period along with placebo.
- Part B-GSK2890457+Liraglutide: Participants with T2D, received oral dose of GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants received liraglutide up to 1.8 mg once daily by subcutaneous injection during the Treatment period along with GSK2890457.
- Part C-Placebo+Metformin: Participants with T2D, received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. Participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2, dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants continued their usual dose of metformin during the treatment period along with placebo, taken one hour prior to placebo as once daily or BID.
- Part C-GSK2890457+Metformin: Participants with T2D, received oral dose of GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5g kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants continued their usual dose of metformin during the treatment period along with GSK2890457, taken one hour prior to GSK2890457 as once daily or BID.
Period: Overall Study
Arm/Group | Part A-Placebo | Part A-GSK2890457 | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Started | 4 | 11 | 6 | 14 | 6 | 12
Completed | 4 | 10 | 6 | 13 | 6 | 12
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A-Placebo: Healthy participants received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. On Day 1 and 42, after overnight fasting, participants received 500 mg IR tablet of metformin just before breakfast. On Day 1 (5 g) and Day 42, matching placebo to GSK2890457 was given in the evening.
- Total: Total of all reporting groups
Arm/Group | Part A-Placebo | Part A-GSK2890457 | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin | Total
Number analyzed (Participants) | 4 | 11 | 6 | 14 | 6 | 12 | 53
Age, Customized [Count of Participants; unit: Participants]
  18 to 70 years | 4 | 11 | 6 | 14 | 6 | 12 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 3 | 4 | 15
  Male | 3 | 10 | 3 | 11 | 3 | 8 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 6 | 1 | 1 | 0 | 2 | 11
  White | 3 | 5 | 5 | 13 | 6 | 10 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE), Serious Adverse Event (SAE) or Death During Part A
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase (ALT) >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalized ratio >1.5.
Time Frame: Up to Follow-up (8 weeks)
Population: All Subjects Population comprised of all randomized participants who received at least one dose of study medication (placebo or GSK2890457).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Participants
  Any AE | 3 | 10
  Any SAE | 0 | 0
  Any Death | 0 | 0

2. Primary Outcome: Number of Participants With Any AE, SAE or Death During Part B and Part C
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as ALT >=3 x ULN, and total bilirubin >=2 x ULN or international normalized ratio >1.5.
Time Frame: Up to Follow-up (8 weeks)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Participants
  Any AE | 1 | 3 | 3 | 3
  Any SAE | 0 | 0 | 0 | 0
  Any Death | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Any Hypoglycemic Events During Part A
Description: Hypoglycemia is defined as symptoms consistent with hypoglycemia (e.g. dizziness, light-headedness, shakiness) which are confirmed by glucometer measurement of complete blood count (CBG) or plasma glucose value of <50 milligram per deciliter (mg/dL) for Part A or <70 mg/dL for Parts B and C (when possible, CBG values were confirmed with a laboratory measurement). In situations when no glucose sample could be measured at the time of the event, the investigator, at his or her discretion, characterized an event as 'hypoglycemia' based on reported signs and symptoms alone. Healthy participant also had asymptomatic blood glucose values <70 mg/dL as a physiological response to altered food intake (e.g., fasting).
Time Frame: Up to Follow-up (8 weeks)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Any Hypoglycemic Events During Part B and Part C
Description: Hypoglycemia is defined as symptoms consistent with hypoglycemia (e.g. dizziness, light-headedness, shakiness) which are confirmed by glucometer measurement of CBG or plasma glucose value of <50 mg/dL for Part A or <70 mg/dL for Parts B and C (when possible, CBG values were confirmed with a laboratory measurement). In situations when no glucose sample could be measured at the time of the event, the investigator, at his or her discretion, characterized an event as 'hypoglycemia' based on reported signs and symptoms alone. Healthy participant also had asymptomatic blood glucose values <70 mg/dL as a physiological response to altered food intake (e.g., fasting).
Time Frame: Up to Follow-up (8 weeks)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part B-Placebo+Liraglutide: Participants with T2D, received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. Participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2, dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants received liraglutide up to 1.8 mg once daily by subcutaneous injection during the Treatment period along with placebo.
- Part C-GSK2890457+Metformin: Participants with T2D, received oral dose of GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5g kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15g to 40g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants continued their usual dose of metformin during the treatment period along with GSK2890457, taken one hour prior to GSK2890457 as once daily or BID.
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Alkaline Phosphatase (ALP), ALT, Aspartate Aminotransferase (AST) and Gamma Glutamyltransferase (GGT) During Double-blind Treatment Period of Part A
Description: The assessments were done pre-dose at Day 1, Day 7, Day 14, Day 28 and Day 42. Baseline value was defined as the assessment done on Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
International unit per liter (IU/L)
  ALP, Day 7 | -6.0 (5.83) | -3.8 (3.28)
  ALP, Day 14 | -1.3 (6.08) | -1.4 (5.30)
  ALP, Day 28: number analyzed (Participants) | 4 | 10
  ALP, Day 28 | 0.0 (4.83) | -1.8 (2.82)
  ALP, Day 42: number analyzed (Participants) | 4 | 10
  ALP, Day 42 | -1.0 (3.37) | -1.8 (4.73)
  ALT, Day 7 | 5.5 (10.15) | -4.1 (6.74)
  ALT, Day 14 | 1.3 (2.99) | -4.4 (8.27)
  ALT, Day 28: number analyzed (Participants) | 4 | 10
  ALT, Day 28 | 2.0 (5.48) | -8.2 (10.76)
  ALT, Day 42: number analyzed (Participants) | 4 | 10
  ALT, Day 42 | 5.3 (17.37) | -7.7 (9.31)
  AST, Day 7 | 2.3 (2.06) | -0.4 (5.73)
  AST, Day 14 | -2.3 (3.40) | 1.4 (5.45)
  AST, Day 28: number analyzed (Participants) | 4 | 10
  AST, Day 28 | -0.8 (3.10) | -3.1 (4.95)
  AST, Day 42: number analyzed (Participants) | 4 | 10
  AST, Day 42 | 2.3 (6.95) | -0.3 (4.62)
  GGT, Day 7 | 1.5 (5.45) | -0.1 (2.39)
  GGT, Day 14 | 1.0 (4.24) | -0.1 (3.27)
  GGT, Day 28: number analyzed (Participants) | 4 | 10
  GGT, Day 28 | 0.8 (4.86) | -2.9 (4.41)
  GGT, Day 42: number analyzed (Participants) | 4 | 10
  GGT, Day 42 | 2.5 (4.36) | -0.5 (3.81)

6. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of ALP, ALT, AST and GGT During the Double-blind Treatment Period of Part B and C
Description: The assessments were done pre-dose at Day -1, Day 7, Day 14, Day 28 and Day 42. Baseline value was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
IU/L
  ALP, Day 7 | 5.3 (11.86) | 5.5 (7.68) | 1.8 (9.62) | -2.2 (9.35)
  ALP, Day 14 | 5.2 (9.45) | 1.8 (5.42) | 6.7 (4.03) | -3.7 (17.92)
  ALP, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  ALP, Day 28 | -0.3 (6.89) | 2.8 (8.88) | 6.3 (15.83) | -2.5 (7.78)
  ALP, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  ALP, Day 42 | 4.3 (8.69) | 2.2 (5.58) | 0.5 (8.50) | -2.8 (9.53)
  ALT, Day 7 | -1.3 (4.84) | -0.1 (3.05) | 1.5 (4.85) | -1.0 (4.61)
  ALT, Day 14 | -2.3 (5.54) | 0.6 (5.75) | 3.0 (10.99) | -6.3 (13.85)
  ALT, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  ALT, Day 28 | -2.5 (4.18) | 0.9 (6.70) | 0.7 (2.80) | -3.8 (9.63)
  ALT, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  ALT, Day 42 | -4.3 (5.13) | 1.0 (10.21) | -0.5 (6.35) | -4.2 (7.79)
  AST, Day 7 | -1.2 (7.39) | 1.1 (2.66) | -0.5 (7.20) | 0.2 (3.04)
  AST, Day 14 | -1.3 (5.96) | 1.9 (3.63) | -1.0 (14.76) | -0.3 (6.02)
  AST, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  AST, Day 28 | -2.0 (4.86) | 2.2 (4.74) | 0.7 (7.61) | 1.4 (4.85)
  AST, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  AST, Day 42 | -3.8 (5.08) | 3.8 (8.19) | 1.0 (4.38) | 1.9 (4.94)
  GGT, Day 7 | 0.7 (0.82) | -1.2 (3.26) | 0.3 (1.97) | 1.3 (3.11)
  GGT, Day 14 | 0.8 (1.33) | -1.4 (5.11) | 5.3 (9.33) | 2.3 (12.74)
  GGT, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  GGT, Day 28 | 0.0 (2.45) | 0.8 (2.80) | 2.3 (5.68) | 0.5 (4.01)
  GGT, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  GGT, Day 42 | -0.7 (2.34) | 0.2 (4.18) | -0.7 (4.55) | -0.9 (4.52)

7. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Electrolytes, Glucose Phosphorus Inorganic and Urea/Blood Urea Nitrogen (BUN) During the Double-blind Treatment Period of Part A
Description: The electrolytes include calcium, chloride, carbon dioxide content/bicarbonate, potassium, magnesium and sodium. Assessments were done pre-dose at on Day 1, Day 7, Day 14, Day 28 and Day 42. Baseline value was defined as the assessment done on Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles (mmol)/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Millimoles (mmol)/L
  Calcium, Day 7 | -0.025 (0.1019) | -0.023 (0.0718)
  Calcium, Day 14 | 0.056 (0.0624) | -0.023 (0.0875)
  Calcium, Day 28: number analyzed (Participants) | 4 | 10
  Calcium, Day 28 | 0.056 (0.0985) | -0.010 (0.0554)
  Calcium, Day 42: number analyzed (Participants) | 4 | 10
  Calcium, Day 42 | 0.050 (0.0611) | -0.022 (0.0729)
  Chloride, Day 7 | 0.8 (2.50) | 1.2 (1.89)
  Chloride, Day 14 | 1.0 (0.82) | 0.4 (1.63)
  Chloride, Day 28: number analyzed (Participants) | 4 | 10
  Chloride, Day 28 | -1.5 (0.58) | 0.5 (2.12)
  Chloride, Day 42: number analyzed (Participants) | 4 | 10
  Chloride, Day 42 | -0.8 (1.26) | 0.4 (2.12)
  Carbon dioxide/Bicarbonate, Day 7 | 0.3 (1.50) | -1.2 (1.72)
  Carbon dioxide/Bicarbonate, Day 14 | -1.0 (2.16) | -1.9 (1.64)
  Carbon dioxide/Bicarbonate, Day 28: number analyzed (Participants) | 4 | 10
  Carbon dioxide/Bicarbonate, Day 28 | -0.5 (2.08) | -1.2 (1.75)
  Carbon dioxide/Bicarbonate, Day 42: number analyzed (Participants) | 4 | 10
  Carbon dioxide/Bicarbonate, Day 42 | -2.5 (2.08) | -2.8 (2.44)
  Glucose, Day 7 | -0.0 (0.51) | -0.1 (0.35)
  Glucose, Day 14 | -0.0 (0.44) | -0.3 (0.37)
  Glucose, Day 28: number analyzed (Participants) | 4 | 10
  Glucose, Day 28 | -0.1 (0.45) | -0.2 (0.33)
  Glucose, Day 42: number analyzed (Participants) | 4 | 10
  Glucose, Day 42 | -0.2 (0.22) | -0.3 (0.28)
  Potassium, Day 7 | 0.15 (0.387) | -0.15 (0.491)
  Potassium, Day 14 | 0.20 (0.804) | -0.15 (0.406)
  Potassium, Day 28: number analyzed (Participants) | 4 | 10
  Potassium, Day 28 | -0.07 (0.419) | -0.13 (0.419)
  Potassium, Day 42: number analyzed (Participants) | 4 | 10
  Potassium, Day 42 | 0.30 (0.673) | -0.16 (0.548)
  Magnesium, Day 7 | -0.0206 (0.05306) | -0.0299 (0.02658)
  Magnesium, Day 14 | -0.0617 (0.07119) | -0.0486 (0.02478)
  Magnesium, Day 28: number analyzed (Participants) | 4 | 10
  Magnesium, Day 28 | -0.0411 (0.05812) | -0.0288 (0.03384)
  Magnesium, Day 42: number analyzed (Participants) | 4 | 10
  Magnesium, Day 42 | -0.0308 (0.02055) | -0.0247 (0.06484)
  Sodium, Day 7 | 0.3 (2.99) | 0.8 (1.60)
  Sodium, Day 14 | -0.3 (1.26) | -0.2 (1.78)
  Sodium, Day 28: number analyzed (Participants) | 4 | 10
  Sodium, Day 28 | 1.0 (3.37) | 1.9 (2.23)
  Sodium, Day 42: number analyzed (Participants) | 4 | 10
  Sodium, Day 42 | -1.3 (2.75) | -0.6 (1.65)
  Urea/BUN, Day 7 | -0.179 (1.4428) | -0.325 (0.7732)
  Urea/BUN, Day 14 | -0.268 (1.1795) | -0.746 (0.6859)
  Urea/BUN, Day 28: number analyzed (Participants) | 4 | 10
  Urea/BUN, Day 28 | -0.536 (1.6098) | -0.643 (1.1264)
  Urea/BUN, Day 42: number analyzed (Participants) | 4 | 10
  Urea/BUN, Day 42 | -0.625 (2.1095) | -0.678 (0.7794)
  Phosphorus inorganic, Day 7 | -0.07 (0.165) | -0.04 (0.090)
  Phosphorus inorganic, Day 14 | -0.14 (0.138) | -0.05 (0.071)
  Phosphorus inorganic, Day 28: number analyzed (Participants) | 4 | 10
  Phosphorus inorganic, Day 28 | -0.02 (0.107) | -0.09 (0.112)
  Phosphorus inorganic, Day 42: number analyzed (Participants) | 4 | 10
  Phosphorus inorganic, Day 42 | 0.01 (0.085) | -0.03 (0.138)

8. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Electrolytes, Glucose Phosphorus Inorganic, BUN and Cholesterol During the Double-blind Treatment Period of Part B and C
Description: The electrolytes include calcium, chloride, carbon dioxide content/bicarbonate, potassium, magnesium and sodium. Assessments were done pre-dose at Day -1, Day 7, Day 14, Day 28 and Day 42. Baseline value was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
mmol/L
  Calcium, Day 7 | 0.083 (0.0604) | 0.053 (0.0763) | 0.025 (0.0879) | -0.004 (0.0991)
  Calcium, Day 14 | 0.050 (0.0985) | 0.041 (0.1079) | 0.067 (0.0700) | 0.017 (0.1215)
  Calcium, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Calcium, Day 28 | 0.021 (0.0677) | 0.046 (0.1063) | 0.004 (0.0695) | 0.035 (0.1352)
  Calcium, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Calcium, Day 42 | -0.025 (0.0523) | -0.040 (0.1168) | -0.071 (0.0533) | -0.056 (0.0775)
  Chloride, Day 7 | -1.5 (1.38) | -1.2 (1.48) | 0.8 (2.93) | 0.4 (1.51)
  Chloride, Day 14 | -0.8 (2.64) | -0.1 (1.96) | 0.5 (2.07) | 0.6 (1.88)
  Chloride, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Chloride, Day 28 | 0.8 (2.79) | 0.2 (1.17) | 1.0 (2.45) | 0.3 (1.50)
  Chloride, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Chloride, Day 42 | -1.0 (2.10) | 0.2 (1.96) | 0.5 (2.35) | 0.3 (0.98)
  Carbon dioxide/Bicarbonate, Day 7 | 0.0 (2.10) | -2.0 (3.53) | -2.0 (2.00) | -0.6 (2.11)
  Carbon dioxide/Bicarbonate, Day 14 | -1.8 (1.94) | -1.9 (3.32) | -2.0 (3.10) | -0.7 (2.42)
  Carbon dioxide/Bicarbonate, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Carbon dioxide/Bicarbonate, Day 28 | -1.0 (2.28) | -0.4 (2.47) | -2.3 (2.34) | -0.3 (2.83)
  Carbon dioxide/Bicarbonate, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Carbon dioxide/Bicarbonate, Day 42 | 0.5 (2.59) | -1.8 (1.91) | -2.8 (2.14) | -1.3 (3.14)
  Glucose, Day 7 | -0.3 (1.32) | 0.3 (3.29) | 0.9 (2.41) | -1.7 (1.86)
  Glucose, Day 14 | -0.1 (1.17) | 0.2 (2.10) | 0.5 (2.06) | -2.2 (2.44)
  Glucose, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Glucose, Day 28 | -0.1 (1.71) | -0.2 (2.31) | 1.5 (2.71) | -2.0 (2.76)
  Glucose, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Glucose, Day 42 | 0.2 (1.06) | -0.1 (2.30) | 1.2 (0.70) | 0.1 (1.62)
  Potassium, Day 7 | 0.33 (0.301) | 0.09 (0.369) | 0.28 (0.264) | 0.06 (0.368)
  Potassium, Day 14 | 0.17 (0.258) | 0.20 (0.353) | 0.17 (0.427) | 0.07 (0.355)
  Potassium, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Potassium, Day 28 | 0.28 (0.172) | 0.08 (0.365) | 0.10 (0.253) | -0.07 (0.352)
  Potassium, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Potassium, Day 42 | -0.05 (0.266) | 0.01 (0.266) | -0.05 (0.302) | 0.08 (0.564)
  Magnesium, Day 7 | 0.0206 (0.05665) | 0.0294 (0.04394) | 0.0206 (0.05034) | -0.0206 (0.08496)
  Magnesium, Day 14 | -0.0206 (0.07236) | 0.0176 (0.06184) | 0.0069 (0.05463) | 0.0206 (0.11153)
  Magnesium, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Magnesium, Day 28 | 0.0274 (0.08879) | 0.0379 (0.08951) | 0.0411 (0.09005) | 0.0240 (0.11284)
  Magnesium, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Magnesium, Day 42 | -0.0137 (0.07197) | 0.0063 (0.06014) | -0.0274 (0.03356) | -0.0171 (0.09349)
  Sodium, Day 7 | 1.2 (2.04) | 0.2 (2.58) | 1.3 (1.51) | 0.8 (1.70)
  Sodium, Day 14 | 1.3 (1.97) | 1.4 (2.98) | 1.5 (1.05) | 1.5 (2.07)
  Sodium, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Sodium, Day 28 | 1.8 (1.94) | 1.7 (2.87) | 1.0 (1.26) | 0.6 (1.16)
  Sodium, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Sodium, Day 42 | 0.5 (0.84) | -0.4 (2.90) | -1.0 (1.79) | -1.0 (2.09)
  Urea/BUN, Day 7 | -0.000 (0.7140) | 0.383 (1.0522) | 0.179 (0.6679) | -0.208 (1.0597)
  Urea/BUN, Day 14 | -0.297 (0.9423) | 0.128 (0.9456) | 0.178 (1.9258) | -0.268 (1.1804)
  Urea/BUN, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Urea/BUN, Day 28 | 0.119 (1.8435) | 0.302 (0.7552) | 0.714 (2.0195) | 0.863 (1.3223)
  Urea/BUN, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Urea/BUN, Day 42 | -0.595 (0.4323) | -0.412 (0.8603) | -0.655 (0.4745) | -0.387 (1.0035)
  Cholesterol, Day 42: number analyzed (Participants) | 1 | 5 | 2 | 2
  Cholesterol, Day 42 | -0.853 (NA) — Only one participant was analyzed at this time point. | -0.103 (0.4579) | -0.052 (0.2560) | -0.155 (0.4389)
  Phosphorus inorganic, Day 7 | 0.10 (0.144) | 0.01 (0.089) | -0.03 (0.186) | 0.01 (0.116)
  Phosphorus inorganic, Day 14: number analyzed (Participants) | 6 | 14 | 5 | 12
  Phosphorus inorganic, Day 14 | 0.01 (0.069) | 0.05 (0.090) | -0.10 (0.193) | 0.03 (0.143)
  Phosphorus inorganic, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Phosphorus inorganic, Day 28 | 0.06 (0.107) | -0.01 (0.162) | -0.12 (0.187) | 0.12 (0.116)
  Phosphorus inorganic, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Phosphorus inorganic, Day 42 | 0.01 (0.053) | -0.04 (0.153) | -0.05 (0.097) | -0.00 (0.094)

9. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles (umol)/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Micromoles (umol)/L
  Direct bilirubin, Day 7 | 0.000 (1.3962) | -0.311 (2.2709)
  Direct bilirubin, Day 14 | 0.428 (0.8550) | -0.466 (1.1058)
  Direct bilirubin, Day 28: number analyzed (Participants) | 4 | 10
  Direct bilirubin, Day 28 | -0.428 (0.8550) | -0.855 (1.6618)
  Direct bilirubin, Day 42: number analyzed (Participants) | 4 | 10
  Direct bilirubin, Day 42 | -0.855 (0.9873) | -0.171 (2.2002)
  Total bilirubin, Day 7 | 0.000 (3.6940) | -0.777 (6.4148)
  Total bilirubin, Day 14 | 0.428 (1.6372) | -0.933 (3.0935)
  Total bilirubin, Day 28: number analyzed (Participants) | 4 | 10
  Total bilirubin, Day 28 | 1.283 (3.7917) | -2.565 (4.1300)
  Total bilirubin, Day 42: number analyzed (Participants) | 4 | 10
  Total bilirubin, Day 42 | 0.855 (2.9618) | 0.513 (5.9264)
  Creatinine, Day 7 | 2.2 (11.12) | -6.4 (6.95)
  Creatinine, Day 14 | -4.4 (11.41) | -4.8 (9.97)
  Creatinine, Day 28: number analyzed (Participants) | 4 | 10
  Creatinine, Day 28 | 0.0 (7.22) | -7.1 (6.97)
  Creatinine, Day 42: number analyzed (Participants) | 4 | 10
  Creatinine, Day 42 | -2.2 (11.12) | -8.8 (4.17)
  Uric acid, Day 7 | -7.4 (43.27) | -10.3 (39.19)
  Uric acid, Day 14 | -14.9 (46.71) | -17.8 (26.60)
  Uric acid, Day 28: number analyzed (Participants) | 4 | 10
  Uric acid, Day 28 | -1.5 (38.05) | 4.2 (56.99)
  Uric acid, Day 42: number analyzed (Participants) | 4 | 10
  Uric acid, Day 42 | -7.4 (35.15) | -26.2 (27.50)

10. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- Part C-Placebo+Metformin: Participants with T2D, received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. Participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2, dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants continued their usual dose of metformin during the treatment period along with placebo as once daily or BID.
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
umol/L
  Direct bilirubin, Day 7 | 0.542 (1.4118) | -0.208 (0.6646) | -0.513 (1.3594) | -0.200 (0.9530)
  Direct bilirubin, Day 14 | 0.314 (0.6876) | -0.305 (0.6578) | -0.086 (0.1431) | -0.185 (0.9379)
  Direct bilirubin, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Direct bilirubin, Day 28 | 0.513 (0.9366) | -0.197 (1.1823) | -0.171 (1.1598) | -0.014 (0.7732)
  Direct bilirubin, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Direct bilirubin, Day 42 | 0.599 (0.8635) | -0.197 (0.5708) | -0.200 (0.7978) | -0.328 (0.6780)
  Total bilirubin, Day 7 | 0.570 (5.9891) | -0.855 (2.2991) | -3.705 (4.8867) | 0.000 (2.5258)
  Total bilirubin, Day 14 | -0.570 (4.1418) | -0.611 (2.2851) | -0.855 (0.9366) | 0.285 (2.5082)
  Total bilirubin, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total bilirubin, Day 28 | -0.000 (3.2445) | 0.132 (3.1578) | -0.855 (5.1584) | 0.998 (2.2424)
  Total bilirubin, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total bilirubin, Day 42 | -1.425 (2.9453) | 0.263 (2.6898) | -0.285 (2.9453) | -0.428 (1.6507)
  Creatinine, Day 7 | 4.6 (6.41) | 3.0 (4.10) | 6.9 (5.60) | 3.4 (4.47)
  Creatinine, Day 14 | -0.1 (3.85) | 4.2 (5.61) | 5.7 (8.21) | 4.6 (6.48)
  Creatinine, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Creatinine, Day 28 | 1.9 (6.38) | 2.0 (4.99) | 4.9 (7.88) | 8.2 (11.05)
  Creatinine, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Creatinine, Day 42 | -1.0 (3.60) | -2.4 (7.48) | 0.6 (3.98) | -0.8 (5.52)
  Uric acid, Day 7 | 15.9 (54.73) | 25.1 (30.26) | 3.0 (52.09) | 9.9 (34.81)
  Uric acid, Day 14 | -11.9 (37.43) | 15.3 (35.74) | -21.8 (55.88) | 25.3 (50.03)
  Uric acid, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Uric acid, Day 28 | 2.0 (61.78) | 16.9 (45.09) | -13.9 (54.60) | 34.7 (41.27)
  Uric acid, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Uric acid, Day 42 | -5.0 (29.96) | 7.8 (38.35) | 9.9 (11.70) | 0.5 (26.78)

11. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Albumin and Total Protein During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
g/L
  Albumin, Day 7 | 0.0 (2.45) | -0.3 (1.90)
  Albumin, Day 14 | 2.0 (1.83) | 0.4 (1.96)
  Albumin, Day 28: number analyzed (Participants) | 4 | 10
  Albumin, Day 28 | 2.5 (2.89) | 0.4 (1.07)
  Albumin, Day 42: number analyzed (Participants) | 4 | 10
  Albumin, Day 42 | 2.5 (2.08) | 0.0 (2.36)
  Total protein, Day 7 | -0.8 (3.77) | -2.1 (3.24)
  Total protein, Day 14 | -0.3 (2.06) | -1.2 (4.00)
  Total protein, Day 28: number analyzed (Participants) | 4 | 10
  Total protein, Day 28 | 1.0 (2.45) | -2.2 (2.74)
  Total protein, Day 42: number analyzed (Participants) | 4 | 10
  Total protein, Day 42 | 0.8 (2.06) | -3.1 (4.25)

12. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Albumin and Total Protein During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
g/L
  Albumin, Day 7 | 2.0 (2.00) | 3.1 (2.11) | 1.3 (2.07) | 0.5 (1.88)
  Albumin, Day 14 | 2.7 (3.01) | 2.6 (2.17) | 0.8 (2.79) | 1.6 (3.15)
  Albumin, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Albumin, Day 28 | 1.8 (1.94) | 2.8 (2.54) | 2.3 (1.97) | 1.9 (2.71)
  Albumin, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Albumin, Day 42 | 0.0 (1.90) | 0.4 (2.02) | -0.8 (1.94) | -1.3 (2.23)
  Total protein, Day 7 | 3.0 (3.03) | 2.9 (2.51) | 1.0 (4.15) | 1.1 (3.12)
  Total protein, Day 14 | 4.0 (5.10) | 2.7 (3.67) | 1.7 (4.72) | 2.2 (4.41)
  Total protein, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total protein, Day 28 | 3.2 (4.17) | 3.2 (3.65) | 2.8 (4.17) | 3.1 (4.03)
  Total protein, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total protein, Day 42 | 0.5 (1.38) | -0.6 (2.79) | -0.7 (3.08) | -1.5 (3.45)

13. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Insulin During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles (pmol)/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Picomoles (pmol)/L
  Day 7: number analyzed (Participants) | 4 | 9
  Day 7 | -1.256 (26.7142) | 12.516 (28.0792)
  Day 14: number analyzed (Participants) | 4 | 8
  Day 14 | 8.072 (32.6673) | 1.973 (13.8798)
  Day 28: number analyzed (Participants) | 4 | 8
  Day 28 | -11.659 (16.5012) | 8.969 (42.2377)
  Day 42: number analyzed (Participants) | 3 | 7
  Day 42 | -22.721 (17.5213) | -13.735 (11.7418)

14. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Insulin During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
pmol/L
  Day 7: number analyzed (Participants) | 5 | 9 | 4 | 10
  Day 7 | -20.21 (33.619) | -20.05 (90.341) | 45.11 (44.635) | -29.59 (41.312)
  Day 14: number analyzed (Participants) | 5 | 9 | 4 | 10
  Day 14 | -21.65 (61.873) | -9.62 (62.083) | -79.39 (33.851) | -41.14 (67.791)
  Day 28: number analyzed (Participants) | 5 | 8 | 4 | 10
  Day 28 | -53.41 (48.574) | -35.18 (76.905) | 34.28 (70.064) | -7.22 (39.675)
  Day 42: number analyzed (Participants) | 5 | 8 | 4 | 9
  Day 42 | -12.99 (40.953) | -8.12 (48.862) | 34.28 (36.025) | 35.28 (61.179)

15. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Amylase and Lipase the Double-blind Treatment Period of Part B of Study
Description: The assessments were done pre-dose at Day -1 and Day 42. Baseline value was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 42) value. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) and Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units (U)/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide
Number analyzed (Participants) | 6 | 14
Units (U)/L
  Amylase, Day 42: number analyzed (Participants) | 6 | 13
  Amylase, Day 42 | 6.0 (10.90) | 9.2 (29.49)
  Lipase, Day 42: number analyzed (Participants) | 6 | 13
  Lipase, Day 42 | 7.5 (21.25) | 18.8 (71.07)

16. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Triiodothyronine (T3) Uptake During the Double-blind Treatment Period of Part B and C
Description: The assessments were done pre-dose at Day -1 and Day 42. Baseline value was defined as the assessment done Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 42) value. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) and Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 5 | 8 | 4 | 10
Ratio | -0.018 (0.0110) | -0.009 (0.0164) | 0.002 (0.0126) | -0.001 (0.0173)

17. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Total Thyroxine and Total T3 During the Double-blind Treatment Period of Part B and C
Description: as for outcome 16
Time Frame: Baseline (Day -1) and Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles (nmol)/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Nanomoles (nmol)/L
  Total thyroxine: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total thyroxine | 0.8578 (7.70771) | 1.0891 (6.62201) | -5.1478 (7.09618) | -2.3597 (8.19189)
  Total T3: number analyzed (Participants) | 1 | 5 | 2 | 2
  Total T3 | -0.3 (NA) — Only one participant was analyzed for this arm at this time point. | 0.1 (0.31) | -0.2 (0.15) | -0.2 (0.16)

18. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters of Thyroid Stimulating Hormone During the Double-blind Treatment Period of Part B and C
Description: The assessments were done pre-dose at Day -1, Day 7 and Day 42. Baseline value was defined as the assessment done Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliunits (mu/L)
Groups:
- Part C-GSK2890457+Metformin: Participants with T2D, received oral dose of GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants continued their usual dose of metformin during the treatment period along with GSK2890457, taken one hour prior to GSK2890457 as once daily or BID.
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Milliunits (mu/L)
  Day 7: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 7 |  | -5.790 (NA) — Only one participant was analyzed for this arm at this time point. |  |
  Day 42 | 0.137 (0.5036) | -0.067 (0.2826) | -0.187 (0.8308) | 0.149 (0.3342)

19. Primary Outcome: Change From Baseline in Hematology Parameters of Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, White Blood Cell (WBC) Count During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells (GI)/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Giga cells (GI)/L
  Basophils, Day 7 | 0.00 (0.000) | 0.00 (0.000)
  Basophils, Day 14 | -0.03 (0.050) | 0.01 (0.030)
  Basophils, Day 28: number analyzed (Participants) | 4 | 10
  Basophils, Day 28 | 0.00 (0.000) | 0.00 (0.000)
  Basophils, Day 42: number analyzed (Participants) | 4 | 10
  Basophils, Day 42 | 0.00 (0.000) | 0.00 (0.000)
  Eosinophils, Day 7 | -0.03 (0.050) | -0.03 (0.065)
  Eosinophils, Day 14 | -0.03 (0.050) | 0.00 (0.063)
  Eosinophils, Day 28: number analyzed (Participants) | 4 | 10
  Eosinophils, Day 28 | 0.10 (0.141) | 0.00 (0.067)
  Eosinophils, Day 42: number analyzed (Participants) | 4 | 10
  Eosinophils, Day 42 | 0.03 (0.050) | 0.00 (0.094)
  Lymphocytes, Day 7 | -0.22 (0.287) | -0.01 (0.644)
  Lymphocytes, Day 14 | -0.22 (0.050) | -0.06 (0.448)
  Lymphocytes, Day 28: number analyzed (Participants) | 4 | 10
  Lymphocytes, Day 28 | -0.23 (0.189) | -0.32 (0.496)
  Lymphocytes, Day 42: number analyzed (Participants) | 4 | 10
  Lymphocytes, Day 42 | 0.15 (0.520) | 0.05 (0.264)
  Monocytes, Day 7 | -0.08 (0.126) | -0.05 (0.104)
  Monocytes, Day 14 | -0.10 (0.000) | -0.05 (0.069)
  Monocytes, Day 28: number analyzed (Participants) | 4 | 10
  Monocytes, Day 28 | -0.05 (0.058) | 0.01 (0.120)
  Monocytes, Day 42: number analyzed (Participants) | 4 | 10
  Monocytes, Day 42 | -0.05 (0.129) | -0.06 (0.052)
  Total Neutrophils, Day 7 | 0.15 (0.947) | 0.02 (0.852)
  Total Neutrophils, Day 14 | 0.50 (0.990) | -0.13 (0.583)
  Total Neutrophils, Day 28: number analyzed (Participants) | 4 | 10
  Total Neutrophils, Day 28 | -0.32 (0.465) | 0.14 (0.841)
  Total Neutrophils, Day 42: number analyzed (Participants) | 4 | 10
  Total Neutrophils, Day 42 | 0.48 (0.556) | -0.01 (0.743)
  Platelet count, Day 7 | -4.8 (26.08) | -1.9 (16.65)
  Platelet count, Day 14 | -14.0 (45.91) | 3.8 (16.30)
  Platelet count, Day 28: number analyzed (Participants) | 4 | 10
  Platelet count, Day 28 | -11.5 (51.98) | 9.7 (29.04)
  Platelet count, Day 42: number analyzed (Participants) | 4 | 10
  Platelet count, Day 42 | -8.8 (17.37) | 3.1 (25.18)
  WBC count, Day 7 | -0.15 (1.310) | -0.11 (1.118)
  WBC count, Day 14 | 0.18 (0.964) | -0.15 (0.715)
  WBC count, Day 28: number analyzed (Participants) | 4 | 10
  WBC count, Day 28 | -0.50 (0.490) | -0.16 (1.047)
  WBC count, Day 42: number analyzed (Participants) | 4 | 10
  WBC count, Day 42 | 0.65 (0.988) | -0.01 (0.984)

20. Primary Outcome: Change From Baseline in Hematology Parameters of Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, WBC Count During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
GI/L
  Basophils, Day 7 | 0.0270 (0.03653) | 0.0047 (0.01481) | 0.0047 (0.00650) | -0.0078 (0.01673)
  Basophils, Day 14 | 0.0037 (0.01122) | 0.0041 (0.01653) | -0.0015 (0.01195) | -0.0066 (0.01893)
  Basophils, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Basophils, Day 28 | -0.0002 (0.01418) | 0.0050 (0.01755) | -0.0065 (0.04654) | -0.0068 (0.02566)
  Basophils, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Basophils, Day 42 | 0.0098 (0.00895) | 0.0019 (0.01499) | -0.0190 (0.04076) | -0.0122 (0.02336)
  Eosinophils, Day 7 | 0.02 (0.040) | 0.04 (0.088) | -0.01 (0.055) | -0.03 (0.054)
  Eosinophils, Day 14 | 0.01 (0.032) | 0.03 (0.086) | -0.02 (0.043) | -0.00 (0.044)
  Eosinophils, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Eosinophils, Day 28 | 0.01 (0.049) | 0.02 (0.083) | 0.01 (0.067) | -0.00 (0.079)
  Eosinophils, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Eosinophils, Day 42 | 0.01 (0.045) | 0.06 (0.128) | -0.02 (0.041) | -0.01 (0.044)
  Lymphocytes, Day 7 | 0.31 (0.333) | 0.11 (0.304) | 0.09 (0.253) | 0.14 (0.511)
  Lymphocytes, Day 14 | 0.18 (0.275) | 0.04 (0.295) | 0.08 (0.280) | 0.18 (0.371)
  Lymphocytes, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Lymphocytes, Day 28 | 0.08 (0.300) | 0.05 (0.631) | 0.05 (0.317) | 0.25 (0.594)
  Lymphocytes, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Lymphocytes, Day 42 | 0.02 (0.158) | -0.11 (0.228) | -0.11 (0.307) | -0.07 (0.364)
  Monocytes, Day 7 | 0.04 (0.109) | -0.01 (0.100) | 0.01 (0.149) | 0.00 (0.115)
  Monocytes, Day 14 | -0.05 (0.125) | -0.04 (0.122) | 0.06 (0.125) | 0.06 (0.096)
  Monocytes, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Monocytes, Day 28 | 0.03 (0.147) | -0.03 (0.080) | 0.06 (0.099) | 0.03 (0.132)
  Monocytes, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Monocytes, Day 42 | 0.00 (0.100) | -0.06 (0.120) | -0.00 (0.087) | -0.03 (0.074)
  Total Neutrophils, Day 7 | 0.27 (0.431) | -0.13 (0.666) | -0.54 (0.500) | 0.38 (0.786)
  Total Neutrophils, Day 14 | 0.38 (0.932) | -0.19 (0.722) | -0.27 (0.591) | 0.64 (0.876)
  Total Neutrophils, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total Neutrophils, Day 28 | -0.01 (0.608) | -0.17 (0.778) | -0.48 (1.097) | 0.36 (1.048)
  Total Neutrophils, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Total Neutrophils, Day 42 | -0.24 (0.404) | -0.14 (0.561) | -0.50 (0.845) | -0.10 (0.645)
  Platelet count, Day 7 | 18.3 (24.21) | 8.9 (18.10) | 5.0 (20.82) | 5.8 (21.36)
  Platelet count, Day 14 | 12.8 (29.31) | 7.0 (11.02) | 1.2 (31.94) | 12.9 (15.97)
  Platelet count, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Platelet count, Day 28 | 4.5 (23.87) | 10.8 (21.90) | 0.5 (34.01) | 10.4 (16.91)
  Platelet count, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Platelet count, Day 42 | -2.0 (23.13) | -13.2 (30.99) | -13.8 (41.97) | -15.3 (28.56)
  WBC count, Day 7 | 0.65 (0.582) | -0.01 (0.791) | -0.43 (0.900) | 0.48 (1.099)
  WBC count, Day 14 | 0.52 (0.997) | -0.17 (0.862) | -0.13 (0.933) | 0.88 (1.131)
  WBC count, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  WBC count, Day 28 | 0.08 (0.728) | -0.13 (1.057) | -0.35 (1.414) | 0.63 (1.643)
  WBC count, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  WBC count, Day 42 | -0.20 (0.533) | -0.26 (0.413) | -0.62 (1.130) | -0.22 (0.824)

21. Primary Outcome: Change From Baseline in Hematology Parameters of Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
g/L
  Hemoglobin, Day 7 | 0.8 (2.06) | -2.0 (6.36)
  Hemoglobin, Day 14 | 4.0 (4.24) | -0.9 (7.30)
  Hemoglobin, Day 28: number analyzed (Participants) | 4 | 10
  Hemoglobin, Day 28 | 11.3 (7.41) | 0.5 (3.84)
  Hemoglobin, Day 42: number analyzed (Participants) | 4 | 10
  Hemoglobin, Day 42 | 9.8 (7.37) | 0.9 (9.34)
  MCHC, Day 7 | 1.8 (2.99) | 5.4 (7.31)
  MCHC, Day 14 | -0.5 (9.40) | 0.0 (5.71)
  MCHC, Day 28: number analyzed (Participants) | 4 | 10
  MCHC, Day 28 | 8.5 (7.55) | 6.3 (6.02)
  MCHC, Day 42: number analyzed (Participants) | 4 | 10
  MCHC, Day 42 | 17.5 (7.19) | 9.0 (11.75)

22. Primary Outcome: Change From Baseline in Hematology Parameters of Hemoglobin and MCHC During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
g/L
  Hemoglobin, Day 7 | 0.2 (5.08) | -1.0 (4.67) | -4.3 (5.85) | -3.4 (6.89)
  Hemoglobin, Day 14 | 0.2 (9.66) | -1.1 (6.50) | 1.7 (4.93) | -2.1 (13.10)
  Hemoglobin, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Hemoglobin, Day 28 | 0.3 (3.98) | -1.1 (7.63) | -1.2 (8.68) | -0.3 (8.70)
  Hemoglobin, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Hemoglobin, Day 42 | 0.0 (2.97) | -0.8 (4.87) | -2.8 (4.58) | -4.8 (5.83)
  MCHC, Day 7 | -2.0 (4.82) | -4.1 (5.40) | -4.5 (2.74) | -2.8 (4.97)
  MCHC, Day 14 | 2.0 (7.21) | -3.8 (5.28) | -1.2 (3.54) | -2.6 (5.09)
  MCHC, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  MCHC, Day 28 | 1.7 (7.15) | -1.9 (4.80) | -2.0 (5.22) | -1.4 (3.53)
  MCHC, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  MCHC, Day 42 | 2.0 (6.16) | 0.2 (4.36) | -0.2 (2.79) | 0.8 (4.63)

23. Primary Outcome: Change From Baseline in Hematology Parameters of Red Blood Cell (RBC) Count and Reticulocytes During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells (TI)/L
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Trillion cells (TI)/L
  RBC count, Day 7 | -0.008 (0.1014) | -0.116 (0.1851)
  RBC count, Day 14 | 0.090 (0.0337) | -0.084 (0.2313)
  RBC count, Day 28: number analyzed (Participants) | 4 | 10
  RBC count, Day 28 | 0.258 (0.1455) | -0.045 (0.1516)
  RBC count, Day 42: number analyzed (Participants) | 4 | 10
  RBC count, Day 42 | 0.107 (0.3192) | -0.115 (0.2632)
  Reticulocytes, Day 7 | 0.0115 (0.00281) | 0.0014 (0.01076)
  Reticulocytes, Day 14 | 0.0077 (0.00189) | -0.0017 (0.01001)
  Reticulocytes, Day 28: number analyzed (Participants) | 4 | 10
  Reticulocytes, Day 28 | 0.0073 (0.00151) | 0.0071 (0.01522)
  Reticulocytes, Day 42: number analyzed (Participants) | 4 | 10
  Reticulocytes, Day 42 | 0.0022 (0.00998) | 0.0044 (0.01396)

24. Primary Outcome: Change From Baseline in Hematology Parameters of RBC Count and Reticulocytes During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: TI/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
TI/L
  RBC count, Day 7 | 0.018 (0.1916) | 0.004 (0.1536) | -0.107 (0.2013) | -0.085 (0.2176)
  RBC count, Day 14 | -0.030 (0.2999) | -0.011 (0.2282) | 0.093 (0.2399) | -0.072 (0.4808)
  RBC count, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  RBC count, Day 28 | 0.002 (0.1229) | -0.023 (0.2500) | 0.020 (0.3651) | -0.003 (0.2871)
  RBC count, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  RBC count, Day 42 | 0.032 (0.0662) | -0.031 (0.1445) | -0.053 (0.1978) | -0.168 (0.1987)
  Reticulocytes, Day 7: number analyzed (Participants) | 5 | 9 | 4 | 10
  Reticulocytes, Day 7 | 0.0020 (0.01123) | -0.0003 (0.01284) | -0.0210 (0.02605) | -0.0015 (0.02719)
  Reticulocytes, Day 14: number analyzed (Participants) | 5 | 9 | 4 | 10
  Reticulocytes, Day 14 | -0.0019 (0.02127) | 0.0095 (0.02126) | -0.0286 (0.02354) | 0.0147 (0.02091)
  Reticulocytes, Day 28: number analyzed (Participants) | 5 | 8 | 4 | 10
  Reticulocytes, Day 28 | 0.0029 (0.01673) | 0.0035 (0.01697) | -0.0304 (0.01024) | -0.0052 (0.01674)
  Reticulocytes, Day 42: number analyzed (Participants) | 5 | 8 | 4 | 10
  Reticulocytes, Day 42 | 0.0062 (0.01283) | 0.0096 (0.01916) | -0.0200 (0.03679) | -0.0042 (0.02667)

25. Primary Outcome: Change From Baseline in Hematology Parameter of Hematocrit During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Ratio
  Day 7 | 0.0000 (0.00365) | -0.0128 (0.01836)
  Day 14 | 0.0128 (0.00943) | -0.0026 (0.01975)
  Day 28: number analyzed (Participants) | 4 | 10
  Day 28 | 0.0228 (0.01921) | -0.0066 (0.01127)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 0.0060 (0.02780) | -0.0089 (0.02614)

26. Primary Outcome: Change From Baseline in Hematology Parameter of Hematocrit During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Ratio
  Day 7 | 0.0032 (0.01240) | 0.0019 (0.01645) | -0.0082 (0.01837) | -0.0072 (0.02007)
  Day 14 | -0.0028 (0.02218) | 0.0011 (0.02030) | 0.0057 (0.01628) | -0.0036 (0.03707)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | -0.0003 (0.00900) | -0.0003 (0.02237) | -0.0010 (0.02832) | 0.0003 (0.02786)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | -0.0022 (0.01032) | -0.0025 (0.01509) | -0.0087 (0.01154) | -0.0159 (0.01827)

27. Primary Outcome: Change From Baseline in Hematology Parameter of Mean Corpuscle Hemoglobin (MCH) During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Picograms
  Day 7 | 0.25 (0.420) | 0.31 (0.589)
  Day 14 | 0.27 (0.881) | 0.32 (0.453)
  Day 28: number analyzed (Participants) | 4 | 10
  Day 28 | 0.70 (0.816) | 0.37 (0.427)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 1.40 (0.841) | 0.89 (0.924)

28. Primary Outcome: Change From Baseline in Hematology Parameter of MCH During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Picograms
  Day 7 | -0.02 (0.160) | -0.21 (0.315) | -0.23 (0.314) | -0.18 (0.434)
  Day 14 | 0.18 (0.319) | -0.10 (0.476) | -0.25 (0.689) | 0.03 (0.454)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | 0.17 (0.484) | 0.01 (0.487) | -0.20 (0.410) | -0.08 (0.343)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | -0.12 (0.412) | 0.08 (0.668) | -0.28 (0.500) | 0.02 (0.333)

29. Primary Outcome: Change From Baseline in Hematology Parameter of Mean Corpuscle Volume (MCV) During the Double-blind Treatment Period of Part A
Description: as for outcome 5
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Femtoliters
  Day 7 | 0.15 (1.323) | -0.55 (0.792)
  Day 14 | 0.85 (1.348) | 0.95 (0.682)
  Day 28: number analyzed (Participants) | 4 | 10
  Day 28 | -0.30 (1.393) | -0.62 (1.105)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | -0.90 (1.219) | 0.35 (1.866)

30. Primary Outcome: Change From Baseline in Hematology Parameter of MCV During the Double-blind Treatment Period of Part B and C
Description: as for outcome 6
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Femtoliters
  Day 7 | 0.35 (1.067) | 0.39 (1.296) | 0.40 (0.443) | 0.25 (1.119)
  Day 14 | 0.02 (0.659) | 0.54 (1.134) | -0.47 (1.544) | 0.76 (1.925)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | 0.05 (0.967) | 0.55 (1.381) | -0.18 (1.465) | 0.17 (1.303)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | -0.90 (1.279) | 0.07 (1.768) | -0.78 (1.468) | -0.27 (1.263)

31. Primary Outcome: Number of Participants With Abnormal Urinalyisis Dipstick and Microscopic Results During the Double-blind Treatment Period of Part A
Description: The assessments were done pre-dose at Day 1, Day 7, Day 14, Day 28 and Day 42. Only those parameters for which at least one value of abnormal urinalysis result was reported are summarized. The participants were categorized as rare, trace, +1, 2+, RBC's and WBC's as <1, 1, 2, 3 and 4. Protein concentration ranged from trace to 1+, where trace indicated lowest concentration and 1+ indicated highest concentration. Trace was the highest concentration for occult blood. Bacteria concentration ranged from rare to moderate, where rare indicated lowest concentration and moderate indicated highest concentration. Ketones ranged from trace to 1+, where trace indicated lowest concentration and 1+ indicated highest concentration. RBC and WBC ranged from <1 to 4, where <1 indicated lowest concentration and 4 indicated highest concentration. Highest concentration indicated worse outcome.
Time Frame: Up to Day 42
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part A-Placebo: Healthy participants received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) prior to breakfast (morning) and 10 g (2 unit) prior to dinner (evening). On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. On Day 1 and 42, after overnight fasting, participants received 500 mg immediate release (IR) tablet of metformin just before breakfast. On Day 1 (5 g) and Day 42, matching placebo to GSK2890457 was given in the evening.
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Participants
  Protein, Trace, Day 1 | 1 | 3
  Protein, Trace, Day 7 | 0 | 2
  Protein, 1+, Day 7 | 0 | 1
  Protein, Trace, Day 14 | 0 | 1
  Protein, Trace, Day 28 | 1 | 4
  Protein, Trace, Day 42 | 2 | 2
  Bacteria, Rare, Day 1 | 1 | 0
  Bacteria, Rare, Day 42 | 0 | 1
  Bacteria, Moderate, Day 42 | 1 | 0
  Occult blood, Trace, Day 1 | 1 | 0
  Occult blood, Trace, Day 14 | 1 | 1
  Occult blood, Trace, Day 28 | 0 | 1
  Ketones, 1+, Day 1 | 1 | 0
  Ketones, 1+, Day 7 | 0 | 1
  Ketones, Trace, Day 14 | 1 | 0
  Ketones, Trace, Day 28 | 1 | 0
  Ketones, Trace, Day 42 | 1 | 0
  RBC's, 1, Day 1 | 1 | 1
  RBC's, 3, Day 1 | 1 | 0
  RBC's, <1, Day 1 | 0 | 1
  RBC's, 1, Day 7 | 0 | 1
  RBC's, <1, Day 7 | 0 | 1
  RBC's, 2, Day 14 | 1 | 0
  RBC's, <1, Day 14 | 0 | 2
  RBC's, 1, Day 28 | 0 | 2
  RBC's, <1, Day 28 | 2 | 2
  RBC's, 1, Day 42 | 0 | 1
  RBC's, 2, Day 42 | 2 | 0
  RBC's, <1, Day 42 | 0 | 1
  WBC's, 1, Day 1 | 2 | 2
  WBC's, <1, Day 1 | 0 | 1
  WBC's, 1, Day 7 | 0 | 2
  WBC's, <1, Day 7 | 0 | 1
  WBC's, 2, Day 14 | 1 | 1
  WBC's, <1, Day 14 | 1 | 1
  WBC's, 1, Day 28 | 2 | 0
  WBC's, <1, Day 28 | 0 | 1
  WBC's, 1, Day 42 | 0 | 1
  WBC's, 2, Day 42 | 1 | 0
  WBC's, 4, Day 42 | 1 | 1

32. Primary Outcome: Number of Participants With Abnormal Urinalyisis Dipstick and Microscopic Results During the Double-blind Treatment Period of Part B
Description: The assessments were done pre-dose at Day -1, Day 7, Day 14, Day 28 and Day 42. Only those parameters for which at least one value of abnormal urinalysis result was reported are summarized. The participants were categorized as few, trace, +1, 2+, 3+, 0-3, 10-20, 0-5, 6-10, and 20-40. Few was the highest concentration of bacteria. Occult blood ranged from trace to 1+, trace indicated lowest and 1+ indicated highest concentration. Epithelial cell ranged from 0-5 to 10-20, 0-5 indicated lowest and 10-20 indicated highest concentration. Glucose ranged from trace to 3+, trace indicated lowest and 3+ indicated highest concentration. 0-5 was highest concentration for hyaline casts. Ketone ranged from trace to 1+, trace indicated lowest and 1+ indicated highest concentration. RBC and WBC ranged from 0-3 to 20-40, 0-3 indicated lowest and 20-40 indicated highest concentration. Highest concentration indicated worse outcome.
Time Frame: Up to Day 42
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide
Number analyzed (Participants) | 6 | 14
Participants
  Bacteria, Few, Day -1 | 1 | 0
  Occult Blood, 1+, Day 14 | 0 | 1
  Occult Blood, Trace, Day 28 | 0 | 1
  Occult Blood, Trace, Day 42 | 0 | 1
  Epithelial Cells, 10-20, Day -1 | 1 | 0
  Epithelial Cells, 0-5, Day 7 | 1 | 1
  Epithelial Cells, 6-10, Day 7 | 1 | 0
  Epithelial Cells, 0-5, Day 14 | 1 | 2
  Epithelial Cells, 0-5, Day 42 | 1 | 1
  Glucose, 1+, Day -1 | 0 | 4
  Glucose, 3+, Day -1 | 0 | 2
  Glucose, Trace, Day -1 | 2 | 1
  Glucose, 1+, Day 7 | 0 | 1
  Glucose, 3+, Day 7 | 1 | 2
  Glucose, Trace, Day 7 | 0 | 3
  Glucose, 1+, Day 14 | 0 | 1
  Glucose, 2+, Day 14 | 0 | 1
  Glucose, 3+, Day 14 | 1 | 1
  Glucose, Trace, Day 14 | 0 | 3
  Glucose, 1+, Day 28 | 0 | 2
  Glucose, 2+, Day 28 | 1 | 1
  Glucose, 3+, Day 28 | 0 | 2
  Glucose, Trace, Day 28 | 0 | 1
  Glucose, 1+, Day 42 | 2 | 0
  Glucose, 2+, Day 42 | 0 | 2
  Glucose, 3+, Day 42 | 0 | 3
  Glucose, Trace, Day 42 | 1 | 3
  Hyaline Casts, 0-5, Day 14 | 1 | 0
  Ketones, 1+, Day 7 | 0 | 1
  Ketones, Trace, Day 14 | 2 | 1
  Ketones, Trace, Day 28 | 0 | 1
  RBC's, 0-3, Day-1 | 1 | 0
  RBC's, 0-3, Day 7 | 1 | 0
  RBC's, 0-3, Day 14 | 0 | 1
  RBC's, 0-3, Day 28 | 0 | 1
  RBC's, 0-3, Day 42 | 0 | 1
  WBC's, 20-40, Day -1 | 1 | 0
  WBC's, 0-5, Day 7 | 1 | 1
  WBC's, 6-10, Day 7 | 1 | 0
  WBC's, 0-5, Day 14 | 1 | 1
  WBC's, 0-5, Day 28 | 0 | 1
  WBC's, 0-5, Day 42 | 1 | 1

33. Primary Outcome: Number of Participants With Abnormal Urinalyisis Dipstick and Microscopic Results During the Double-blind Treatment Period of Part C
Description: The assessments were done pre-dose at Day -1, Day 7, Day 14, Day 28 and Day 42. The participants were categorized as few, many, moderate, trace, +1, 2+, 3+, 0-3, 10-20, 0-5, 6-10, 20-40, 40-60. Protein and ketone ranged from trace to 1+, trace indicated lowest and 1+ indicated highest concentration. Bacteria and uric acid crystals ranged from few to moderate, few indicated lowest and moderate indicated highest concentration. Trace was the highest concentration of occult blood. Epithelial cells ranged from 0-5 to >10, 0-5 indicated lowest and >10 indicated highest concentration. Glucose ranged from trace to 3+, trace indicated lowest and 3+ indicated highest concentration. 0-1 was highest concentration for hyaline casts. RBC and WBC ranged from 0-3 to 40-60, 0-3 indicated lowest and 20-40 indicated highest concentration. Highest concentration indicated worse outcome.
Time Frame: Up to Day 42
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 12
Participants
  Protein, 1+, Day 7 | 0 | 1
  Protein, Trace, Day 7 | 0 | 2
  Protein, Trace, Day 14 | 1 | 1
  Protein, 1+, Day 28 | 0 | 1
  Bacteria, Few, Day -1 | 0 | 1
  Bacteria, Many, Day -1 | 1 | 0
  Bacteria, Few, Day 7 | 0 | 4
  Bacteria, Many, Day 7 | 1 | 0
  Bacteria, Many, Day 14 | 0 | 1
  Bacteria, Moderate, Day 14 | 1 | 0
  Bacteria, Few, Day 28 | 1 | 1
  Bacteria, Many, Day 28 | 1 | 0
  Bacteria, Many, Day 42 | 1 | 0
  Bacteria, Moderate, Day 42 | 0 | 1
  Occult Blood, Trace, Day 42 | 0 | 1
  Epithelial Cells, 0-10, Day -1 | 0 | 1
  Epithelial Cells, 0-10, Day 7 | 0 | 1
  Epithelial Cells, 0-5, Day 7 | 0 | 1
  Epithelial Cells, 6-10, Day 7 | 0 | 1
  Epithelial Cells, 0-5, Day 14 | 0 | 1
  Epithelial Cells, >10, Day 14 | 0 | 1
  Epithelial Cells, 0-10, Day 28 | 1 | 1
  Epithelial Cells, 0-10, Day 42 | 0 | 1
  Glucose, 1+, Day -1 | 0 | 1
  Glucose, 2+, Day -1 | 0 | 1
  Glucose, 3+, Day -1 | 0 | 6
  Glucose, 1+, Day 7 | 1 | 0
  Glucose, 2+, Day 7 | 0 | 2
  Glucose, 3+, Day 7 | 1 | 1
  Glucose, Trace, Day 7 | 1 | 2
  Glucose, 1+, Day 14 | 1 | 2
  Glucose, 3+, Day 14 | 0 | 2
  Glucose, Trace, Day 14 | 0 | 4
  Glucose, 2+, Day 28 | 1 | 2
  Glucose, 3+, Day 28 | 1 | 1
  Glucose, Trace, Day 28 | 0 | 2
  Glucose, 1+, Day 42 | 3 | 2
  Glucose, 2+, Day 42 | 0 | 1
  Glucose, 3+, Day 42 | 0 | 4
  Glucose, Trace, Day 42 | 0 | 1
  Hyaline Casts, 0-1, Day 7 | 0 | 1
  Ketones, 1+, Day 7 | 0 | 1
  Ketones, Trace, Day 7 | 0 | 2
  Ketones, Trace, Day 14 | 1 | 1
  Ketones, Trace, Day 28 | 1 | 1
  RBC's, 0-3, Day -1 | 0 | 1
  RBC's, 0-3, Day 7 | 0 | 2
  RBC's, 0-3, Day 14 | 0 | 2
  RBC's, 0-3, Day 28 | 1 | 1
  RBC's, 0-3, Day 42 | 0 | 1
  Uric acid crystals, Moderate, Day 7 | 0 | 1
  Uric acid crystals, Few, Day 14 | 0 | 1
  WBC's, 0-5, Day -1 | 1 | 1
  WBC's, 0-5, Day 7 | 1 | 3
  WBC's, 6-10, Day 7 | 0 | 1
  WBC's, 0-5, Day 14 | 1 | 2
  WBC's, 0-5, Day 28 | 1 | 1
  WBC's, 40-60, Day 28 | 1 | 0
  WBC's, 6-10, Day 42 | 1 | 1

34. Primary Outcome: Mean Specific Gravity Values of Urine During the Double-blind Treatment Period of Part A
Description: Urinary specific gravity is a measure of the concentration of solutes in urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine. The assessments were done pre-dose at Da y 1, Day 7, Day 14, Day 28 and Day 42.
Time Frame: Up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Ratio
  Day 1 | 1.0193 (0.00903) | 1.0175 (0.00794)
  Day 7 | 1.0133 (0.00685) | 1.0165 (0.00887)
  Day 14 | 1.0153 (0.00591) | 1.0152 (0.00752)
  Day 28: number analyzed (Participants) | 4 | 10
  Day 28 | 1.0125 (0.00705) | 1.0122 (0.00983)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 1.0155 (0.00759) | 1.0161 (0.00827)

35. Primary Outcome: Mean Specific Gravity Values of Urine During the Double-blind Treatment Period of Part B and C
Description: Urinary specific gravity is a measure of the concentration of solutes in urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine. The assessments were done pre-dose at Day -1, Day 7, Day 14, Day 28 and Day 42.
Time Frame: Up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Ratio
  Day -1 | 1.0168 (0.00773) | 1.0174 (0.00482) | 1.0172 (0.00627) | 1.0187 (0.00796)
  Day 7 | 1.0208 (0.00794) | 1.0191 (0.00734) | 1.0197 (0.00356) | 1.0208 (0.00688)
  Day 14 | 1.0202 (0.00861) | 1.0196 (0.00812) | 1.0198 (0.00382) | 1.0201 (0.00629)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | 1.0232 (0.00906) | 1.0239 (0.00533) | 1.0213 (0.00505) | 1.0213 (0.00559)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | 1.0137 (0.00535) | 1.0188 (0.00910) | 1.0110 (0.00544) | 1.0172 (0.01021)

36. Primary Outcome: Mean pH Values of Urine During the Double-blind Treatment Period of Part A
Description: Urinalysis parameter included urine pH. pH was calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral. The assessments were done pre-dose on Day 1, Day 7, Day 14, Day 28 and Day 42.
Time Frame: up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
pH
  Day 1 | 5.25 (0.289) | 5.95 (0.472)
  Day 7 | 5.88 (0.854) | 5.86 (0.745)
  Day 14 | 5.50 (0.408) | 5.91 (0.735)
  Day 28: number analyzed (Participants) | 4 | 10
  Day 28 | 6.13 (1.031) | 6.05 (0.832)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 5.63 (0.250) | 6.20 (0.632)

37. Primary Outcome: Mean pH Values of Urine During the Double-blind Treatment Period of Part B and C
Description: Urinalysis parameter included urine pH. pH was calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral. The assessments were done pre-dose on Day -1, Day 7, Day 14, Day 28 and Day 42.
Time Frame: Up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Part C-GSK2890457+Metformin: Participants with T2D, received oral dose of GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 1 5g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) in morning and 10 g (2 unit) in evening. On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. Participants continued their usual dose of metformin during the treatment period along with GSK2890457, taken one hour prior to GSK2890457 as once daily or BID.
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
pH
  Day -1 | 5.92 (0.376) | 6.25 (0.470) | 5.67 (0.408) | 5.83 (0.537)
  Day 7 | 5.83 (0.683) | 5.89 (0.350) | 5.83 (0.816) | 5.42 (0.359)
  Day 14 | 5.67 (0.408) | 6.07 (0.646) | 5.67 (0.516) | 5.63 (0.433)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | 5.75 (0.418) | 5.96 (0.477) | 5.67 (0.408) | 5.63 (0.311)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | 6.00 (0.316) | 6.08 (0.449) | 5.58 (0.376) | 5.58 (0.417)

38. Primary Outcome: Change From Baseline in Vital Sign Parameter of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) During the Double-blind Treatment Period of Part A
Description: Vital sign assessments were performed after resting in a supine or semi-supine position for at least 10 minutes. The assessments were done pre-dose at Day 1, Day 7, Day 14, Day 28 and Day 42. Baseline value was defined as the assessment done on Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Millimeters of mercury (mmHg)
  SBP, Day 7 | 0.8 (11.70) | -4.0 (4.94)
  SBP, Day 14 | -0.5 (1.91) | -3.9 (6.45)
  SBP, Day 28: number analyzed (Participants) | 4 | 10
  SBP, Day 28 | -3.3 (6.45) | -5.5 (7.55)
  SBP, Day 42: number analyzed (Participants) | 4 | 10
  SBP, Day 42 | -1.0 (11.28) | -7.5 (6.19)
  DBP, Day 7 | -5.3 (4.50) | -6.2 (4.12)
  DBP, Day 14 | -1.8 (3.95) | -5.0 (8.51)
  DBP, Day 28: number analyzed (Participants) | 4 | 10
  DBP, Day 28 | -1.3 (5.56) | -8.4 (5.72)
  DBP, Day 42: number analyzed (Participants) | 4 | 10
  DBP, Day 42 | -0.8 (3.30) | -6.4 (7.21)

39. Primary Outcome: Change From Baseline in Vital Sign Parameter of SBP and DBP During the Double-blind Treatment Period of Part B and C
Description: Vital sign assessments were performed after resting in a supine or semi-supine position for at least 10 minutes. The assessments were done pre-dose at Day -1, Day 7, Day 14, Day 28 and Day 42. Baseline value was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
mmHg
  SBP, Day 7 | 1.6 (11.11) | 2.0 (11.05) | 3.2 (6.94) | -3.7 (12.40)
  SBP, Day 14 | 5.6 (9.70) | 3.6 (8.52) | 3.2 (9.28) | -2.8 (9.45)
  SBP, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  SBP, Day 28 | -0.6 (7.43) | 0.2 (9.51) | 4.5 (13.29) | -7.4 (9.62)
  SBP, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  SBP, Day 42 | -2.6 (6.18) | 0.1 (4.31) | 0.0 (10.11) | -3.0 (10.04)
  DBP, Day 7 | -2.4 (6.00) | 0.4 (4.88) | 0.9 (4.53) | -0.8 (5.71)
  DBP, Day 14 | 2.1 (6.87) | 0.8 (3.23) | -0.8 (2.42) | -2.5 (5.70)
  DBP, Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  DBP, Day 28 | -3.3 (3.96) | 0.4 (5.33) | -0.4 (6.06) | -3.4 (5.33)
  DBP, Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  DBP, Day 42 | -1.5 (4.60) | 0.8 (4.32) | 1.1 (4.35) | -3.2 (5.30)

40. Primary Outcome: Change From Baseline in Vital Sign Parameter of Heart Rate (HR) During the Double-blind Treatment Period of Part A
Description: as for outcome 38
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Beats per minute
  Day 7 | 8.0 (6.83) | 4.6 (6.13)
  Day 14: number analyzed (Participants) | 4 | 9
  Day 14 | 6.3 (7.27) | 0.6 (6.75)
  Day 28: number analyzed (Participants) | 4 | 9
  Day 28 | 5.5 (9.57) | 3.3 (7.07)
  Day 42: number analyzed (Participants) | 4 | 9
  Day 42 | -1.3 (7.37) | -4.4 (6.29)

41. Primary Outcome: Change From Baseline in Vital Sign Parameter of HR During the Double-blind Treatment Period of Part B and C
Description: as for outcome 39
Time Frame: Baseline (Day -1) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Beats per minute
  Day 7 | -3.6 (6.37) | 0.3 (7.91) | 0.1 (5.90) | 1.6 (6.81)
  Day 14 | -3.3 (6.65) | 0.4 (7.65) | 0.8 (7.71) | 3.6 (5.72)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | -7.8 (7.37) | 3.7 (7.92) | 1.8 (4.98) | 1.5 (8.70)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | -4.8 (4.45) | 1.6 (7.42) | -3.2 (5.85) | 0.5 (4.75)

42. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Intervals During Part A
Description: Single 12-lead ECGs was obtained after participants rested in a supine position for at least 10 minutes using an ECG machine that automatically calculated the HR and measured PR, QRS, QT, QT duration corrected for HR by Fridericia's formula (QTcF) and QT duration corrected for HR by Bazett's formula (QTcB intervals. The assessments were done at Day 1 (pre-dose, triplicate), Day 42 (pre-dose) and Follow-up Visit. Baseline value was defined as the average of the triplicate pre-dose assessments done on Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 42 and Follow-up) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day 1, Randomization) up to Follow-up (Day 56)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Milliseconds
  PR Interval, Day 42: number analyzed (Participants) | 4 | 10
  PR Interval, Day 42 | 6.3 (11.00) | 1.1 (8.20)
  PR Interval, Follow-up | 9.0 (10.26) | 1.5 (8.30)
  QRS Duration, Day 42: number analyzed (Participants) | 4 | 10
  QRS Duration, Day 42 | 2.2 (3.91) | -2.1 (3.10)
  QRS Duration, Follow-up | 3.9 (6.05) | -0.7 (6.40)
  QT Interval, Day 42: number analyzed (Participants) | 4 | 10
  QT Interval, Day 42 | 10.8 (13.52) | 16.4 (20.32)
  QT Interval, Follow-up | 0.3 (19.29) | -10.2 (12.81)
  QTcB, Day 42: number analyzed (Participants) | 4 | 10
  QTcB, Day 42 | 8.2 (14.56) | -3.3 (14.89)
  QTcB, Follow-up | 6.9 (9.50) | 6.3 (15.65)
  QTcF, Day 42: number analyzed (Participants) | 4 | 10
  QTcF, Day 42 | 9.1 (12.61) | 3.2 (11.85)
  QTcF, Follow-up | 4.8 (7.81) | 0.7 (11.34)

43. Primary Outcome: Change From Baseline in ECG Intervals During Part B and C
Description: Single 12-lead ECGs was obtained after participants rested in a supine position for at least 10 minutes using an ECG machine that automatically calculated the HR and measured PR, QRS, QT, QTcB, QTcF and RR intervals. The assessments were done at Day -1 (pre-dose, triplicate), Day 42 (pre-dose) and Follow-up Visit. Baseline value was defined as the average of the triplicate pre-dose assessments done on Day -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 42 and Follow-up) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -1) up to Follow-up (Day 56)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 13 | 6 | 12
Milliseconds
  PR Interval, Day 42 | 5.56 (6.206) | 3.08 (14.104) | -6.44 (8.334) | -4.44 (10.156)
  PR Interval, Follow-up | -1.11 (14.327) | -3.69 (11.708) | -3.11 (5.652) | -6.28 (13.676)
  QRS Duration, Day 42 | 0.78 (3.897) | -2.62 (3.049) | 0.11 (4.204) | -1.06 (2.947)
  QRS Duration, Follow-up | 0.11 (2.903) | -1.69 (5.985) | 0.78 (1.760) | 0.11 (3.421)
  QT Interval, Day 42 | 8.11 (10.477) | -1.69 (17.212) | 2.78 (17.711) | 0.78 (15.431)
  QT Interval, Follow-up | 1.44 (27.022) | -5.69 (25.885) | 0.78 (7.559) | -5.56 (17.220)
  QTcB, Day 42 | -2.87 (12.081) | -1.51 (14.358) | 0.43 (13.099) | -4.23 (11.896)
  QTcB, Follow-up | -5.89 (7.088) | -10.95 (14.939) | -3.20 (15.699) | -2.14 (17.641)
  QTcF, Day 42 | 1.17 (9.777) | -1.49 (11.971) | 1.22 (7.799) | -2.58 (10.229)
  QTcF, Follow-up | -3.17 (11.117) | -9.10 (12.639) | -1.78 (9.340) | -3.50 (13.849)
  RR Interval, Day 42 | 0.04 (0.045) | -0.00 (0.086) | 0.01 (0.120) | 0.02 (0.074)
  RR Interval, Follow-up | 0.03 (0.107) | 0.02 (0.127) | 0.02 (0.091) | -0.01 (0.088)

44. Primary Outcome: Change From Baseline in the Overall Gastrointestinal (GI) Symptoms Rating Scale (GSRS) Score During the Double-blind Treatment Period of Part A
Description: The impact of GI symptoms on health-related quality of life was assessed using the GSRS. The GSRS is a 15-item related to abdominal pain, reflux, indigestion, diarrhea and constipation syndromes, self-administered questionnaire that assesses the impact of gastrointestinal symptoms during the past week on a scale from 1 (no discomfort at all) to 7 (very severe discomfort). Overall GSRS was the mean of items 1 to 15. Possible overall scores range from 1 to 7, with lower scores indicating a better quality of life with respect to GI symptoms and higher scores indicating a lower quality of life with respect to GI symptoms. Baseline was defined as the assessment done on Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, 14 and 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day 1, Randomization) up to Day 42
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Scores on scale
  Day 7 | 0.02 (0.033) | 0.08 (0.120)
  Day 14 | 0.08 (0.100) | 0.04 (0.105)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 0.02 (0.033) | -0.02 (0.071)

45. Primary Outcome: Change From Baseline in the Overall GSRS Score During the Double-blind Treatment Period of Part B and C
Description: The impact of GI symptoms on health-related quality of life was assessed using the GSRS. The GSRS is a 15-item related to abdominal pain, reflux, indigestion, diarrhea and constipation syndromes, self-administered questionnaire that assesses the impact of gastrointestinal symptoms during the past week on a scale from 1 (no discomfort at all) to 7 (very severe discomfort). Overall GSRS was the mean of items 1 to 15. Possible overall scores range from 1 to 7, with lower scores indicating a better quality of life with respect to GI symptoms and higher scores indicating a lower quality of life with respect to GI symptoms. Baseline was defined as the assessment done on Day -2. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, 14, 28 and 41) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing.
Time Frame: Baseline (Day -2) up to Day 41
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Scores on scale
  Day 7 | 0.03 (0.516) | -0.03 (0.473) | 0.24 (0.397) | 0.13 (0.197)
  Day 14 | -0.09 (0.167) | 0.05 (0.440) | 0.20 (0.386) | 0.28 (0.366)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | -0.21 (0.191) | 0.03 (0.428) | 0.14 (0.281) | 0.27 (0.436)
  Day 41: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 41 | -0.11 (0.259) | -0.12 (0.290) | 0.02 (0.091) | 0.10 (0.325)

46. Primary Outcome: Change From Baseline in In-clinic Body Weight During the Double-blind Treatment Period of Part B and C
Description: During the assessment of body weight in the unit, the participant wore lightweight indoor clothing and removed shoes. The assessments were done pre-dose at Day -1, Day 1, Day 7, Day 14, Day 28, Day 42 and Day 43. Baseline value was defined as the average of Day -1 and Day 1 values. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing. Day 42 value was the average of Day 42 and Day 43 values.
Time Frame: Baseline (Day -1 and Day 1) up to Day 42
Population: Pharmacodynamic (PD) Population comprised of all participants in the All Subjects Population who had Baseline and at least one post-Baseline assessment of the endpoint. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Kilograms (kg)
  Day 7 | -0.12 (0.938) | 0.20 (1.368) | 0.28 (0.579) | 0.47 (0.840)
  Day 14 | 0.37 (1.157) | 0.05 (1.292) | 0.61 (1.009) | 0.56 (0.779)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | 0.15 (1.161) | 0.47 (1.627) | 0.52 (0.612) | 0.27 (1.265)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | -0.74 (1.020) | -0.39 (1.687) | -0.47 (1.104) | 0.42 (1.221)
Statistical Analysis 1: Comparison: Part B-Placebo+Liraglutide vs Part B-GSK2890457+Liraglutide; Part B-Placebo+Liraglutide versus Part B-GSK2890457+Liraglutide for Day 42 change from Baseline in body weight; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Repeated measures analysis of variance was used with terms for treatment, visit, treatment by visit interaction and Baseline; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.38 to 1.75] — Point estimate was calculated as difference in least squares means: Part B-GSK2890457+Liraglutide minus Part B-Placebo+Liraglutide
Statistical Analysis 2: Comparison: Part C-Placebo+Metformin vs Part C-GSK2890457+Metformin; Part C-Placebo+Metformin versus Part C-GSK2890457+Metformin for Day 42 change from Baseline in body weight; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; [statistical method as in outcome 46, analysis 1]; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [-0.20 to 2.36] — Point estimate was calculated as difference in least squares means: Part C-GSK2890457+Metformin minus Part C-Placebo+Metformin

47. Primary Outcome: Percent Change From Baseline in In-clinic Body Weight During the Double-blind Treatment Period of Part B and C
Description: During the assessment of body weight in the unit, the participant wore lightweight indoor clothing and removed shoes. The assessments were done pre-dose at Day -1, Day 1, Day 7, Day 14, Day 28, Day 42 and Day 43. Baseline value was defined as the average of Day -1 and Day 1 values. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Day 7, Day 14, Day 28 and Day 42) values. Percent change was calculated by multiplying the change from Baseline value with 100. If either the Baseline or post-Baseline value was missing, the change from Baseline was set to be missing. Day 42 value was the average of Day 42 and Day 43 values.
Time Frame: Baseline (Day -1 and Day 1) up to Day 42
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
Percent change
  Day 7 | -0.16 (1.020) | 0.18 (1.521) | 0.36 (0.719) | 0.59 (0.892)
  Day 14 | 0.47 (1.252) | -0.04 (1.442) | 0.79 (1.346) | 0.60 (0.780)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | 0.25 (1.264) | 0.39 (1.792) | 0.66 (0.813) | 0.30 (1.371)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | -0.80 (1.199) | -0.51 (1.884) | -0.53 (1.504) | 0.50 (1.365)
Statistical Analysis 1: Comparison: Part B-Placebo+Liraglutide vs Part B-GSK2890457+Liraglutide; Part B-Placebo+Liraglutide versus Part B-GSK2890457+Liraglutide for Day 42 percent change from Baseline in body weight; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; [statistical method as in outcome 46, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-1.64 to 1.87] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: Part C-Placebo+Metformin vs Part C-GSK2890457+Metformin; Part C-Placebo+Metformin versus Part C-GSK2890457+Metformin for Day 42 percent change from Baseline in body weight; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; [statistical method as in outcome 46, analysis 1]; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [-0.24 to 2.75] — [estimate comment as in outcome 46, analysis 2]

48. Primary Outcome: Change From Baseline in Weighted Mean Glucose Area Under the Curves From Time 0 to 24 Hours (AUC [0-24 Hours]) During the Double-blind Treatment Period of Part B and C
Description: AUC was calculated using the linear trapezoid method that is the sum of the areas between each chronological pair of assessments at the time points (at Day -1 and Day 42). The weighted mean was then calculated by dividing the AUC by the length of the time interval over which it was calculated. Baseline was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline (Day -1) values from the post-Baseline value (Day 42). Data is reported for weighted mean glucose AUC (0-4 hour) post-breakfast and AUC (0-24 hour) post-breakfast. Adjusted mean is reported as least square (LS) mean.
Time Frame: Baseline (Day -1) and Day 42
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 13 | 6 | 12
mmol/L
  AUC (0-4 hour) | 0.018 (0.583) | -0.164 (0.390) | 1.194 (0.518) | 0.341 (0.359)
  AUC (0-24 hour) | -0.613 (0.410) | -0.968 (0.278) | 1.376 (0.459) | 0.156 (0.316)
Statistical Analysis 1: Comparison: Part B-Placebo+Liraglutide vs Part B-GSK2890457+Liraglutide; Part B-Placebo+Liraglutide versus Part B-GSK2890457+Liraglutide for Day 42 change from Baseline in AUC (0-4 hour) weighted mean glucose; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -0.182, 95% CI 2-sided [-1.694 to 1.331] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: Part B-Placebo+Liraglutide vs Part B-GSK2890457+Liraglutide; Part B-Placebo+Liraglutide versus Part B-GSK2890457+Liraglutide for Day 42 change from Baseline in AUC (0-24 hour) weighted mean glucose; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -0.356, 95% CI 2-sided [-1.409 to 0.698] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 3: Comparison: Part C-Placebo+Metformin vs Part C-GSK2890457+Metformin; Part C-Placebo+Metformin versus Part C-GSK2890457+Metformin for Day 42 change from Baseline in AUC (0-4 hour) weighted mean glucose; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -0.853, 95% CI 2-sided [-2.232 to 0.526] — [estimate comment as in outcome 46, analysis 2]
Statistical Analysis 4: Comparison: Part C-Placebo+Metformin vs Part C-GSK2890457+Metformin; Part C-Placebo+Metformin versus Part C-GSK2890457+Metformin for Day 42 change from Baseline in AUC (0-24 hour) weighted mean glucose; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -1.219, 95% CI 2-sided [-2.447 to 0.009] — [estimate comment as in outcome 46, analysis 2]

49. Primary Outcome: Change From Baseline in Fasting Glucose During the Double-blind Treatment Period of Part B and C
Description: Baseline was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline (Day -1) values from the post-Baseline value (Day 42). Adjusted mean is reported as LS mean.
Time Frame: Baseline (Day -1) and Day 42 of Part B and C
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 13 | 6 | 12
mmol/L | -0.384 (0.556) | -0.230 (0.375) | 0.136 (0.520) | -0.387 (0.351)
Statistical Analysis 1: Comparison: Part B-Placebo+Liraglutide vs Part B-GSK2890457+Liraglutide; Part B-Placebo+Liraglutide versus Part B-GSK2890457+Liraglutide for Day 42 change from Baseline in fasting glucose; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = 0.155, 95% CI 2-sided [-1.277 to 1.587] — Point estimate was calculated as difference in least squares means: Part B-GSK2890457+Liraglutide minus Part B -Placebo+Liraglutide
Statistical Analysis 2: Comparison: Part C-Placebo+Metformin vs Part C-GSK2890457+Metformin; Part C-Placebo+Metformin versus Part C-GSK2890457+Metformin for Day 42 change from Baseline in fasting glucose; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -0.524, 95% CI 2-sided [-1.939 to 0.892] — [estimate comment as in outcome 46, analysis 2]

50. Primary Outcome: Change From Baseline in Fasting Insulin and Weighted Mean Insulin AUC (0-4 Hour) and AUC (0-24 Hour) During the Double-blind Treatment Period of Part B and C
Description: Two fasting samples 5 minutes apart were taken for insulin. Baseline insulin level was the average of the 2 fasting samples. For insulin weighted mean AUC (0-4 hour) and weighted mean AUC (0-24 hour) was calculated for Baseline (Day -1) and end of treatment (Day 42). AUC was calculated using the linear trapezoid method that is the sum of the areas between each chronological pair of assessments at the time points (at Day -1 and Day 42). The weighted mean was then calculated by dividing the AUC by the length of the time interval over which it was calculated. Baseline was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline (Day -1) values from the post-Baseline value (Day 42). Data is reported for weighted mean insulin AUC (0-4 hour) post-breakfast and AUC (0-24 hour) post-breakfast.
Time Frame: Baseline (Day -1) and Day 42
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 13 | 6 | 12
pmol/L
  Fasting Insulin | -4.887 (16.5321) | 1.133 (20.2106) | -11.946 (28.0383) | 12.300 (45.8067)
  Insulin Weighted Mean AUC 0-4 hour | 69.635 (31.8542) | 14.589 (67.3782) | 57.887 (74.4685) | 10.322 (81.6157)
  Insulin Weighted Mean AUC 0-24 hour | 1.626 (50.3186) | -13.905 (42.6248) | 22.740 (50.2234) | 17.134 (79.9432)

51. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) During the Double-blind Treatment Period of Part B and C
Description: as for outcome 49
Time Frame: Baseline (Day -1) and Day 42
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent of TL hemoglobin
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 13 | 6 | 12
Percent of TL hemoglobin | -0.214 (0.167) | -0.278 (0.113) | 0.018 (0.264) | -0.201 (0.187)
Statistical Analysis 1: Comparison: Part B-Placebo+Liraglutide vs Part B-GSK2890457+Liraglutide; Part B-Placebo+Liraglutide versus Part B-GSK2890457+Liraglutide for Day 42 change from Baseline in HbA1c; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -0.065, 95% CI 2-sided [-0.495 to 0.365] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: Part C-Placebo+Metformin vs Part C-GSK2890457+Metformin; Part C-Placebo+Metformin versus Part C-GSK2890457+Metformin for Day 42 change from Baseline in HbA1c; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; ANCOVA; Terms for treatment and Baseline were included in the model; Mean Difference (Final Values) = -0.219, 95% CI 2-sided [-0.910 to 0.472] — Point estimate was calculated as difference in least squares means: Part C-GSK2890457+Metformin minus Part Part C-Placebo+Metformin

52. Primary Outcome: Change From Baseline in Homeostasis Model of Assessment-Insulin Resistance (HOMA-IR]) During the Double-blind Treatment Period of Part B and C
Description: HOMA-IR was calculated from the Day -1 and Day 42 fasting glucose and insulin values using dataset generated from the HOMA-2 model. It contained the estimates for HOMA-% insulin sensitivity (S) for pairs of fasting glucose and fasting insulin values. Study data was merged with the HOMA dataset by glucose and insulin. HOMA-IR was calculated as 100/HOMA-%S. HOMA-IR was not determined for any values outside the ranges of plasma glucose 3.5 to 25.0 mmol/L (63 - 450 mg/dL) and plasma insulin 20 to 400 pmol/L. Baseline was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline (Day -1) values from the post-Baseline value (Day 42). Data for Part C of the study was not collected because fasting glucose and insulin were not available at the specified time points.
Time Frame: Baseline (Day -1) and Day 42
Population: PD Population. Only those participants available at the specified time points were analyzed. Data for Part C of the study was not collected because fasting glucose and insulin were not available at the specified time points.
Measure: Mean (Standard Deviation); unit: mU*mmol/L^2
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 12 | 0 | 0
mU*mmol/L^2 | -0.150 (0.4970) | 0.017 (0.7222) |  |

53. Primary Outcome: Change From Baseline in Matsuda Index During the Double Blind-treatment Period of Part B and C
Description: The matsuda index was calculated from the Day -1 and Day 42 glucose and insulin results as 10,000 divided by (fasting plasma glucose x fasting plasma insulin x mean glucose at 0-2 hour post-dose x mean insulin at 0-2 hour post dose)^1/2, where glucose was measured in mmol/L and insulin in pmol/L. Baseline was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline (Day -1) values from the post-Baseline value (Day 42). Data for Part C of the study was not collected because fasting glucose and insulin were not available at the specified time points.
Time Frame: Baseline (Day -1) and Day 42
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: Deciliter*mL/mg*mU
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 13 | 0 | 0
Deciliter*mL/mg*mU | -0.991 (0.6904) | -0.602 (2.4187) |  |

54. Primary Outcome: Change From Baseline in Fasting Plasma Glucose (Safety Laboratory) Values During the Double-blind Treatment Period of Part B and C
Description: The assessments were done at Day -1, Day 7, Day 14, Day 28, Day 42 and Follow-up Visit. Baseline was defined as the assessment done on Day -1. Change from Baseline was calculated by subtracting the Baseline (Day -1) values from the post-Baseline (Day 7, 14, 28, 42 and Follow-up visit) values.
Time Frame: Baseline (Day -1) up to Follow-up (Day 56)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 6 | 14 | 6 | 12
mmol/L
  Day 7 | -0.278 (1.3178) | 0.285 (3.2948) | 0.879 (2.4090) | -1.665 (1.8607)
  Day 14 | -0.093 (1.1748) | 0.210 (2.0999) | 0.518 (2.0551) | -2.216 (2.4434)
  Day 28: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 28 | -0.111 (1.7135) | -0.201 (2.3145) | 1.536 (2.7121) | -1.989 (2.7612)
  Day 42: number analyzed (Participants) | 6 | 13 | 6 | 12
  Day 42 | 0.194 (1.0630) | -0.098 (2.2967) | 1.184 (0.6983) | 0.074 (1.6151)
  Follow-up: number analyzed (Participants) | 6 | 13 | 6 | 12
  Follow-up | 0.962 (1.9719) | 0.444 (3.0739) | 1.249 (1.9061) | -1.226 (1.3623)

55. Secondary Outcome: Area Under Plasma Concentration From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-t]) of Liraglutide During the Double-blind Treatment Period of Part B
Description: Blood samples were collected on Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post dose. The AUC (0-t) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. The analysis population included Liraglutide Pharmacokinetic (PK) Population in Part B comprising of all participants in All Subjects Population for whom a PK sample was obtained and analyzed for Liraglutide.
Time Frame: Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4, 5.5, 6, 8, 10, 11.5, 12, 14 and 24 hours post-dose
Population: Liraglutide Pharmacokinetic (PK) Population in Part B. Only those participants available at specified time points were analyzed. Results from descriptive summary used Liraglutide PK Population. However, results of statistical analysis compared Day 42 to Day -1 PK in GSK2890457+Liraglutide group who were in the Liraglutide PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms/mL
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide
Number analyzed (Participants) | 6 | 14
Hour*nanograms/mL
  Day -1: number analyzed (Participants) | 6 | 12
  Day -1 | 2210.15 (74.900) | 1268.65 (91.758)
  Day 42: number analyzed (Participants) | 5 | 11
  Day 42 | 2505.23 (99.731) | 1265.92 (79.435)
Statistical Analysis 1: Comparison: Part B-GSK2890457+Liraglutide; Comparison of Day 42 to Day -1 in GSK2890457+Liraglutide treated participants in the Liraglutide PK Population; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; Mixed Models Analysis; The PK parameter was log-transformed prior to analysis; Ratio = 1.0460, 90% CI 2-sided [0.7290 to 1.5008] — The difference in least squares means and corresponding confidence interval were back-transformed to form ratio of geometric least squares means (Day 42/ Day -1) and confidence interval

56. Secondary Outcome: Maximum Observed Concentration (Cmax) of Liraglutide During the Double-blind Treatment Period of Part B
Description: Blood samples were collected on Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post-dose. The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: as for outcome 55
Population: Liraglutide PK Population in Part B. Only those participants available at the specified time points were analyzed. Results from descriptive summary used Liraglutide PK Population. However, results of statistical analysis compared Day 42 to Day -1 PK in GSK2890457+Liraglutide group who were in the Liraglutide PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/mL
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide
Number analyzed (Participants) | 6 | 14
Nanograms/mL
  Day -1: number analyzed (Participants) | 6 | 12
  Day -1 | 120.00 (66.845) | 72.24 (70.492)
  Day 42: number analyzed (Participants) | 5 | 11
  Day 42 | 128.57 (86.860) | 70.86 (63.525)
Statistical Analysis 1: Comparison: Part B-GSK2890457+Liraglutide; Comparison of Day 42 to Day -1 in GSK2890457+Liraglutide treated participants in the Liraglutide PK Population; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; Mixed Models Analysis; The PK parameter was log-transformed prior to analysis; Ratio = 1.0334, 90% CI 2-sided [0.7810 to 1.3673] — [estimate comment as in outcome 55, analysis 1]

57. Secondary Outcome: Time of Occurrence of Cmax (Tmax) of Liraglutide During the Double-blind Treatment Period of Part B
Description: Blood samples were collected on Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post-dose. The time at which Cmax was observed was determined directly from the raw concentration-time data.
Time Frame: as for outcome 55
Population: Liraglutide PK Population in Part B. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide
Number analyzed (Participants) | 6 | 14
Hours
  Day -1: number analyzed (Participants) | 6 | 12
  Day -1 | 9.74 [2.0 to 11.5] | 8.00 [0.0 to 11.5]
  Day 42: number analyzed (Participants) | 5 | 11
  Day 42 | 9.92 [2.1 to 11.5] | 9.98 [0.8 to 23.8]

58. Secondary Outcome: AUC of Metformin From Time 0 to 10 Hours Post-dose (AUC [0-10 Hour]) During the Double-blind Treatment Period of Part A
Description: Blood samples were collected on Day 1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8 and 10 (pre-dinner) hours post-dose. The AUC (0-10 hour) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. The analysis population included Metformin PK Population in Part A comprising of all participants in All Subjects Population for whom a PK sample was obtained and analyzed for metformin.
Time Frame: Day 1 and Day 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4, 5.5, 6, 8 and 10 hours post-dose
Population: Metformin PK Population in Part A. Only those participants available at specified time points were analyzed. The results from the descriptive summary used the PK Population. However, the results of the statistical analysis compared Day 42 to Day 1 PK only in the GSK2890457 group who were in the PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms/mL
Groups:
- Part A-Placebo: Healthy participants received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID for 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) prior to breakfast (morning) and 10 g (2 unit) prior to dinner (evening). On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. On Day 1 and 42, after overnight fasting, participants received 500 mg IR tablet of metformin just before breakfast. On Day 1 (5 g) and Day 42, matching placebo to GSK2890457 was given in the evening.
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Hour*nanograms/mL
  Day 1 | 4346.8 (19.1) | 3402.6 (26.4)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 5081.9 (21.1) | 2231.7 (38.6)
Statistical Analysis 1: Comparison: Part A-GSK2890457; Comparison of Day 42 to Day 1 in GSK2890457 treated participants in the PK Population; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; Mixed Models Analysis; The PK parameter was log-transformed prior to analysis; Ratio = 0.675, 90% CI 2-sided [0.585 to 0.779] — The difference in least squares means and corresponding confidence interval were back-transformed to form ratio of geometric least squares means (Day 42/ Day 1) and confidence interval

59. Secondary Outcome: Cmax of Metformin During the Double-blind Treatment Period of Part A
Description: Blood samples were collected on Day 1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8 and 10 (pre-dinner) hours post-dose. The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: Day 1 and Day 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4, 5.5, 6, 8 and 10 hours post-dose
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/mL
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Nanograms/mL
  Day 1 | 681.8 (19.0) | 576.2 (24.4)
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 860.1 (18.8) | 374.1 (31.2)
Statistical Analysis 1: Comparison: Part A-GSK2890457; Comparison of Day 42 to Day 1 in GSK2890457 treated participants in the PK Population; Test type: Other — The analysis used an Estimation approach. No hypothesis testing was performed; Mixed Models Analysis; The PK parameter was log-transformed prior to analysis; Ratio = 0.662, 90% CI 2-sided [0.578 to 0.757] — [estimate comment as in outcome 58, analysis 1]

60. Secondary Outcome: Tmax of Metformin During the Double-blind Treatment Period of Part A
Description: Blood samples were collected on Day 1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8 and 10 (pre-dinner) hours post-dose. The time at which Cmax was observed was determined directly from the raw concentration-time data.
Time Frame: Day 1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4, 5.5, 6, 8 and 10 hours post-dose
Population: Metformin PK Population in Part A. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Placebo | Part A-GSK2890457
Number analyzed (Participants) | 4 | 11
Hours
  Day 1 | 3.010 [2.00 to 4.03] | 2.000 [1.00 to 4.00]
  Day 42: number analyzed (Participants) | 4 | 10
  Day 42 | 4.000 [2.00 to 4.03] | 2.000 [2.00 to 5.50]

61. Secondary Outcome: AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-t]) of Metformin During the Double-blind Treatment Period of Part C
Description: Blood samples were planned to be collected on Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post-dose. The AUC 0-t was planned to be determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. The data for PK parameters of metformin during Part C was not collected due to variations in formulation and regimen.
Time Frame: Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post-dose
Population: Metformin PK Population in Part C comprised of all participants in the All Subjects Population for whom a PK sample was obtained and analyzed for metformin. The data for PK parameters of metformin during Part C was not collected due to variations in formulation and regimen.
Arm/Group | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 0 | 0

62. Secondary Outcome: Cmax of Metformin During the Double-blind Treatment Period of Part C
Description: Blood samples were planned to be collected on Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post-dose. The first occurrence of the Cmax was planned to be determined directly from the raw concentration-time data. The data for PK parameters of metformin during Part C was not collected due to variations in formulation and regimen.
Time Frame: as for outcome 61
Population: Metformin PK Population in Part C. The data for PK parameters of metformin during Part C was not collected due to variations in formulation and regimen.
Arm/Group | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Tmax of Metformin During the Double-blind Treatment Period of Part C
Description: Blood samples were planned to be collected on Day -1 and 42 at pre-dose (0 hour), 15 minutes, 30 minutes, 1, 1.5, 2, 4 (pre-lunch), 5.5, 6, 8, 10 (pre-dinner), 11.5, 12, 14 and 24 hours post-dose. The time at which Cmax was observed was planned to be determined directly from the raw concentration-time data. The data for PK parameters of metformin during Part C was not collected due to variations in formulation and regimen.
Time Frame: as for outcome 61
Population: as for outcome 62
Arm/Group | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected up to Follow-up (8 weeks).
Description: All Subjects Population was used.
Groups:
- Part A-Placebo: Healthy participants received oral dose of matching placebo to GSK2890457 as units of 5 g kit BID or 6 weeks. Each unit of 5 g placebo kit contained 3 sachets of powder and a bottle containing 3 capsules. The powder was mixed with 12 ounces of flavored water, capsules were taken with 120-240 mL of water. The participants were titrated up from 15 g to 40 g over a 7 day period, if tolerated. On Day 2 the dose was 15 g, taken 5 g (1 unit) prior to breakfast (morning) and 10 g (2 unit) prior to dinner (evening). On Day 4, 15 g (3 unit doses) in morning and 15 g (3 unit doses) in evening. On Day 7, 20 g (4 unit doses) in morning and 20 g (4 unit doses) in evening. On Day 1 and 42, after overnight fasting, participants received 500 mg IR tablet of metformin just before breakfast. On Day 1 (5 g) and Day 42, matching placebo to GSK2890457 was given in the evening.
Arm/Group | Part A-Placebo | Part A-GSK2890457 | Part B-Placebo+Liraglutide | Part B-GSK2890457+Liraglutide | Part C-Placebo+Metformin | Part C-GSK2890457+Metformin
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/11 | 0/6 | 0/14 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/11 | 0/6 | 0/14 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 3/4 | 10/11 | 1/6 | 3/14 | 3/6 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-Placebo (N=4) | Part A-GSK2890457 (N=11) | Part B-Placebo+Liraglutide (N=6) | Part B-GSK2890457+Liraglutide (N=14) | Part C-Placebo+Metformin (N=6) | Part C-GSK2890457+Metformin (N=12)
Flatulence (Gastrointestinal disorders) | 2 | 9 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 5 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0
Claustrophobia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.